CLINICAL TRIAL: NCT05004181
Title: A Phase II Trial to Evaluate the Safety and Immunogenicity of SARS-CoV-2 Monovalent and Multivalent RNA-based Vaccines in Healthy Subjects
Brief Title: Safety and Immunogenicity of RNA-based Vaccines Against SARS-CoV-2 Variants in Healthy Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BNT162-17; 2021-003458-22 (EudraCT Number)
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: SARS-CoV-2 Infection; COVID-19; SARS-CoV-2 Acute Respiratory Disease; SARS (Disease)
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Disease | interventions — BNT162 Vaccine; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part A - Cohort 1: 18 to 55 years of age (Experimental): Participants received 1 dose of BNT162b2 (B.1.1.7 + B.1.617.2) of 30 µg.
  Interventions: Biological: Multivalent BNT162b2 (B.1.1.7 + B.1.617.2)
- Part A - Cohort 2: 18 to 55 years of age (Experimental): Participants received 2 doses of BNT162b2 (B.1.1.7 + B.1.617.2) of 30 µg.
  Interventions: Biological: Multivalent BNT162b2 (B.1.1.7 + B.1.617.2)
- Part A - Cohort 3: 18 to 55 years of age (Experimental): Participants received1 dose of BNT162b2 (B.1.1.7) of 30 µg.
  Interventions: Biological: Monovalent BNT162b2 (B.1.1.7)
- Part A - Cohort 4: 18 to 55 years of age (Experimental): Participants received 1 dose of BNT162b2 (B.1.617.2) of 30 µg.
  Interventions: Biological: Monovalent BNT162b2 (B.1.617.2)
- Part A - Cohort 5: 18 to 55 years of age (Experimental): Participants received 1 dose of BNT162b2 of 30 µg.
  Interventions: Biological: BNT162b2
- Part A - Cohort 6: 18 to 55 years of age (Experimental): Participants received 3 doses of BNT162b2 (B.1.1.7 + B.1.617.2) of 30 µg.
  Interventions: Biological: Multivalent BNT162b2 (B.1.1.7 + B.1.617.2)
- Part B - Cohort 1: 18 to 85 years of age (Experimental): Participants received 1 dose of BNT162b2 (B.1.1.7 + B.1.617.2) of 30 µg.
  Interventions: Biological: Multivalent BNT162b2 (B.1.1.7 + B.1.617.2)
- Part B - Cohort 4: 18 to 85 years of age (Experimental): Participants received 1 dose of BNT162b2 (B.1.617.2) of 30 µg.
  Interventions: Biological: Monovalent BNT162b2 (B.1.617.2)
- Part B - Cohort 6: 18 to 85 years of age (Experimental): Participants received 3 doses of BNT162b2 (B.1.1.7 + B.1.617.2) of 30 µg.
  Interventions: Biological: Multivalent BNT162b2 (B.1.1.7 + B.1.617.2)
- Part C - Cohort 7: 18 to 85 years of age (Experimental): Participants received 1 dose of BNT162b2 (B.1.1.529.1) of 30 µg.
  Interventions: Biological: Monovalent BNT162b2 (B.1.1.529.1)
- Part C - Cohort 8: 18 to 85 years of age (Experimental): Participants received 1 dose of BNT162b2 of 30 µg.
  Interventions: Biological: BNT162b2
- Part C - Cohort 9: 18 to 85 years of age (Other): Participants received no vaccination within 3 months after Visit 1.
  Interventions: Other: Observational

INTERVENTIONS:
Biological: BNT162b2 — Intramuscular (IM)
  Arms: Part A - Cohort 5: 18 to 55 years of age; Part C - Cohort 8: 18 to 85 years of age
Biological: Multivalent BNT162b2 (B.1.1.7 + B.1.617.2) — Intramuscular (IM)
  Arms: Part A - Cohort 1: 18 to 55 years of age; Part A - Cohort 2: 18 to 55 years of age; Part A - Cohort 6: 18 to 55 years of age; Part B - Cohort 1: 18 to 85 years of age; Part B - Cohort 6: 18 to 85 years of age
Biological: Monovalent BNT162b2 (B.1.1.7) — Intramuscular (IM)
  Arms: Part A - Cohort 3: 18 to 55 years of age
Biological: Monovalent BNT162b2 (B.1.617.2) — Intramuscular (IM)
  Arms: Part A - Cohort 4: 18 to 55 years of age; Part B - Cohort 4: 18 to 85 years of age
Biological: Monovalent BNT162b2 (B.1.1.529.1) — Intramuscular (IM)
  Arms: Part C - Cohort 7: 18 to 85 years of age
Other: Observational — No vaccination within 3 months after Visit 1.
  Arms: Part C - Cohort 9: 18 to 85 years of age

SUMMARY:
This trial consisted of three parts, Part A, Part B, and Part C, and evaluated the safety and immunogenicity of a third (booster) injection of the multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2), and the safety and immunogenicity of a third booster injection of the monovalent vaccine BNT162b2 (B.1.617.2) or BNT162b2 (B.1.1.7), in participants who had received two doses of the parent vaccine BNT162b2 at 30 µg, at least 6 months after the second dose of BNT162b2. It also evaluated the safety and immunogenicity of a three-dose regimen of BNT162b2 (B.1.1.7 + B.1.617.2) in participants who had not received prior Coronavirus Disease 2019 (COVID-19) vaccination. In addition, the safety and immunogenicity of BNT162b2 (B.1.1.529.1) or BNT162b2 given as a third or fourth vaccine dose to RNA COVID-19 vaccine-experienced participants with history of SARS-CoV-2 Omicron variant infection was evaluated and contrasted with the natural immune response reached after infection with the SARS-CoV-2 Omicron variant in RNA COVID-19 vaccine-experienced participants.

DETAILED DESCRIPTION:
Trial participants in Part A were assigned to one of 6 cohorts (Cohort 1-6). Trial participants in Part B were assigned to one of 3 cohorts (Cohort 1, 4, and 6). Trial participants in Part C were randomized in a 2:2:1 ratio into 3 cohorts (Cohort 7-9).

ELIGIBILITY:
Inclusion Criteria:

* Had given informed consent by signing the informed consent form (ICF) before initiation of any trial-specific procedures.
* Volunteers who at the time of consent were:
* Part A: 18 to 55 years old.
* Part B and Part C: 18 to 85 years old (~60% should be 18 to 55 years old and ~40% 56 to 85 years old).
* For Cohorts 1 to 5: In Part A, who had received BNT162b2 vaccine (30 µg, two-dose regimen) in either a clinical trial or as part of the governmental vaccination programs at least 6 months before Visit 0. Participants who were currently enrolled in the Phase III BNT162-02 / C4591001 (NCT04368728) trial, had already been unblinded, and had previously received two doses of BNT162b2 at least 6 months earlier could be included (for Cohorts 1 and 4 in Part B, prior enrollment and dosing in the C4591001 trial was mandatory). At enrollment into Part B of this trial, their participation in the C4591001 trial was terminated. Participants should have not had experienced COVID-19 based on medical history.
* For Cohort 6: Were COVID-19 vaccine-naïve and had not experienced COVID-19 based on their medical history.
* Were willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, and other trial procedures.
* Were overall healthy at Visit 0 in the clinical judgment of the investigator based on the medical history, clinical assessment (including physical examination, vital signs, blood and urine clinical laboratory tests, 12-lead electrocardiogram (ECG), and oral swab for Nucleic Acid Amplification-based Test (NAAT)-based Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) testing).
* Note: Healthy volunteers with pre-existing stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 12 weeks before Visit 0, could be included.
* Note: Volunteers who had hepatitis C (HCV) infection, but had completed curative treatment based on the medical history could be included. Volunteers who had or have hepatitis B (HBV) or human immunodeficiency virus (HIV) based on the medical history could not be included.
* Agreed not to enroll in another trial of an Investigational Medicinal Product (IMP), starting after Visit 0 and continuously until the last planned visit in this trial.
* Women of childbearing potential (WOCBP) had to test negative in a urine beta-human chorionic gonadotropin (β-HCG) test at Visits 0 and 1.
* WOCBP had to agree to practice a highly effective form of contraception starting at Visit 0 and continuously until 28 days after their last IMP administration in this trial.
* WOCBP had to confirm that they practiced an acceptable form of contraception for the 14 days prior to Visit 0.
* WOCBP had to agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction starting after Visit 0 and continuously until 28 days after their last IMP injection in this trial.
* Men who are sexually active with a WOCBP and had not had a vasectomy had to agree to use a highly effective form of contraception with their female partner of childbearing potential starting after Visit 0 and continuously until 28 days after their last IMP injection in this trial.
* Men had to be willing to refrain from sperm donation, starting after Visit 0 and continuously until 28 days after their last vaccination.
* For Part C, Cohorts 7, 8, and 9: Had received two or three documented doses of any authorized COVID-19 RNA-based vaccine (e.g., BNT162b2 [Comirnaty] or the Moderna vaccine [Spikevax]) prior to being diagnosed with SARS-CoV-2 infection from January 2022 onwards (and limited to a period when there was a high prevalence of SARS-CoV-2 Omicron infections).
* Note: The interval between the last COVID-19 RNA-based vaccine administered and randomization should have been >4 months. The latest prior diagnosed SARS-CoV-2 infection should have been at least 2 months before randomization. The latest SARS-CoV-2 infection should have been documented with a result from a NAAT (as a preferable option). In case no historic NAAT result was available proving prior SARS-CoV-2 infection, the local positive result of SARS-CoV-2 N-binding antibodies done at screening was sufficient.

Exclusion Criteria:

* Any existing condition which could have affected vaccine injection and/or assessment of local reactions assessment, e.g., tattoos, severe scars, etc.
* Any bleeding diathesis or condition associated with prolonged bleeding that could have, in the opinion of the investigator, contraindicated intramuscular injection.
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that, in the investigator's judgment, made the participant inappropriate for the trial.
* Any current febrile illness (body temperature ≥38.0°C/≥100.4°F) or other acute illness within 48 h prior to Day 1/IMP injection in this trial.
* Any current or history of cardiovascular diseases, e.g., myocarditis, pericarditis, myocardial infarction, congestive heart failure, cardiomyopathy or clinically significant arrhythmias, unless such disease was not considered relevant for participation in this trial in the investigator's judgment.
* History of COVID-19 and/or clinical (based on COVID-19 symptoms/signs alone, if a SARS CoV 2 NAAT result was not available) or microbiological (based on COVID-19 symptoms/signs and a positive SARS CoV 2 NAAT result) evidence of prior infection with SARS CoV 2 at screening (Visit 0).
* Note: not applicable for Part C.
* History of Guillain-Barré syndrome.
* Known or suspected immunodeficiency.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g., anaphylaxis) to any component of the trial IMPs.
* History or known allergy, hypersensitivity, or intolerance to the trial IMP including any excipients of the IMPs in this trial.
* Had received any SARS CoV 2 vaccination other than BNT162b2 (30 µg BNT162b2 given as a course of two doses approximately 21 days apart).
* Note: not applicable for Part C.
* Had received a live or live attenuated vaccine within 28 days prior to Day 1/IMP injection.
* Had received any other vaccines within 14 days before or after any IMP injection, e.g., influenza, tetanus, pneumococcal, hepatitis A or B. When possible standard of care vaccinations should been planned with the trial IMP administrations in mind.
* Individuals who received treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids (if systemic corticosteroids were administered for ≥14 days at a dose of ≥20 mg/day of prednisone or equivalent), e.g., for cancer or an autoimmune disease, or planned receipt throughout this trial. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids were permitted.
* Receipt of blood/plasma products or immunoglobulin, from 60 days before IMP administration or planned receipt throughout this trial.
* Participation in other trials involving IMP within 28 days or 5 half-lives (whichever was longer) prior to Visit 1 and/or during trial participation, besides participation in trials with BNT162b2.
* Were pregnant or breastfeeding or are planning pregnancy within 28 days after last IMP treatment.
* Were vulnerable individuals as per International Conference on Harmonisation (ICH) E6 definition, i.e., are individuals whose willingness to volunteer in a clinical trial may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate.
* For Part C, Cohorts 7, 8, and 9: Vaccination with other non-RNA or unauthorized COVID-19 vaccines.
* For Part C, Cohorts 7, 8, and 9: Vaccination with any COVID-19 vaccine after SARS-CoV-2 infection from January 2022 onwards (and limited to a period when there was a high prevalence of SARS-CoV-2 Omicron infections).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1380 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (35):
- United States (14):
  - Collaborative Neuroscience Network LLC, Long Beach, California
  - California Research Foundation, San Diego, California
  - Clinical Research Consulting, Llc, Milford, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - Medpharmics, LLC, Gulfport, Mississippi
  - Amici Clinical Research, Warren Township, New Jersey
  - Rochester Clinical Research, Rochester, New York
  - Aventiv Research Inc., Columbus, Ohio
  - ARC Clinical Research, Austin, Texas
  - North Texas Infectious Diseases Consultants, Dallas, Texas
  - Clinical Trials of Texas Inc., San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
- Germany (4):
  - CRS Clinical Research Services Berlin, Berlin
  - IKF Institut fuer klinische Forschung Frankfurt, Frankfurt am Main
  - CRS Clinical Research Services Mannheim GmbH, Mannheim
  - Studienzentrum Brinkum Dr. Lars Pohlmeier und Torsten Drescher, Stuhr
- South Africa (12):
  - JOSHA Research, Bloemfontein, Free State
  - Langeberg Medicross Medical Centre, Kraaifontein, Western Cape
  - Paarl Research Centre, Paarl, Western Cape
  - Synexus Helderberg Clinical Trial Centre, Somerset West, Western Cape
  - Worthwhile Clinical Trials, Benoni
  - Tiervlei Trial Centre, Cape Town
  - Midrand Medical Centre, Halfway House
  - Newtown Clinical Research, Johannesburg
  - Global Clinical Trials, Pretoria
  - Botho ke Bontle Health Service, Pretoria
  - Synexus SA Stanza Clinical Research Centre, Pretoria
  - Jongaie Research, Medicross Pretoria West, Pretoria
- Turkey (Türkiye) (5):
  - Ankara University Faculty of Medicine, Avicenna Hospital, Ankara
  - Hacettepe University Hospital, Ankara
  - Bagcilar Medipol Mega University Hospital, Istanbul
  - Istanbul University Medical Faculty, Istanbul
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muik A, Quandt J, Lui BG, Bacher M, Lutz S, Grunenthal M, Toker A, Grosser J, Ozhelvaci O, Blokhina O, Shpyro S, Vogler I, Salisch N, Tureci O, Sahin U. Immunity against conserved epitopes dominates after two consecutive exposures to SARS-CoV-2 Omicron BA.1. Cell Rep. 2024 Aug 27;43(8):114567. doi: 10.1016/j.celrep.2024.114567. Epub 2024 Aug 3. PMID 39097927
- [Derived] Muik A, Lui BG, Quandt J, Diao H, Fu Y, Bacher M, Gordon J, Toker A, Grosser J, Ozhelvaci O, Grikscheit K, Hoehl S, Kohmer N, Lustig Y, Regev-Yochay G, Ciesek S, Beguir K, Poran A, Vogler I, Tureci O, Sahin U. Progressive loss of conserved spike protein neutralizing antibody sites in Omicron sublineages is balanced by preserved T cell immunity. Cell Rep. 2023 Aug 29;42(8):112888. doi: 10.1016/j.celrep.2023.112888. Epub 2023 Jul 31. PMID 37527039
- [Derived] Muik A, Lui BG, Bacher M, Wallisch AK, Toker A, Couto CIC, Guler A, Mampilli V, Schmitt GJ, Mottl J, Ziegenhals T, Fesser S, Reinholz J, Wernig F, Schraut KG, Hefesha H, Cai H, Yang Q, Walzer KC, Grosser J, Strauss S, Finlayson A, Kruger K, Ozhelvaci O, Grikscheit K, Kohmer N, Ciesek S, Swanson KA, Vogel AB, Tureci O, Sahin U. Exposure to BA.4/5 S protein drives neutralization of Omicron BA.1, BA.2, BA.2.12.1, and BA.4/5 in vaccine-experienced humans and mice. Sci Immunol. 2022 Dec 23;7(78):eade9888. doi: 10.1126/sciimmunol.ade9888. Epub 2022 Dec 23. PMID 36378074

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult male and female participants were eligible if they had received two doses of the parent vaccine BNT162b2 at 30 µg, and the second dose of BNT162b2 was at least 6 months ago (Part A Cohorts 1 to 5, Part B Cohorts 1 and 4), or had not received prior Coronavirus Disease 2019 (COVID-19) vaccination (Part A Cohort 6, Part B Cohort 6) or had received 2 or 3 injections of any authorized COVID-19 RNA-based vaccine and were subsequently diagnosed with SARS-CoV-2 infection from January 2022 onwards
Groups:
- Part A - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2); Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2): Participants received 1 dose of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2) as a single injection on Day 1
- Part A - Cohort 2: 2 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2): Participants received 2 doses of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2) as a single injection one on Day 1 and one on Day 56
- Part A - Cohort 3: 1 Dose of 30 μg BNT162b2 (B.1.1.7): Participants received 1 dose of 30 μg monovalent vaccine BNT162b2 (B.1.1.7) on Day 1
- Part A - Cohort 4: 1 Dose of 30 μg BNT162b2 (B.1.617.2); Part B - Cohort 4: 1 Dose 30 μg BNT162b2 (B.1.617.2): Participants received 1 dose of 30 μg monovalent vaccine BNT162b2 (B.1.617.2) on Day 1
- Part A - Cohort 5: 1 Dose of 30 μg BNT162b2 (Original Vaccine); Part C - Cohort 8: 1 Dose of 30 μg BNT162b2 (Original Vaccine): Participants received 1 dose of 30 μg BNT162b2 original vaccine on Day 1
- Part A - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2); Part B - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2): Participants received 3 doses of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2), as a single injection one on Day 1, one on Day 21 and one approximately 6 months after the second dose
- Part C - Cohort 7: 1 Dose of 30 μg BNT162b2 (B.1.1.529): Participants received 1 dose of 30 μg monovalent vaccine BNT162b2 (B.1.1.529) on Day 1
- Part C - Cohort 9: No Vaccination: No vaccination was given to Cohort 9 participants within 3 months after Visit 1. After the 3-month follow-up period, subjects in Cohort 9 were to be offered a BNT162b2 vaccination, depending on the epidemiological situation, local regulatory authority recommendations, and/or variant vaccine authorization status.
Period: Overall Study
Arm/Group | Part A - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 2: 2 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 3: 1 Dose of 30 μg BNT162b2 (B.1.1.7) | Part A - Cohort 4: 1 Dose of 30 μg BNT162b2 (B.1.617.2) | Part A - Cohort 5: 1 Dose of 30 μg BNT162b2 (Original Vaccine) | Part A - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part B - Cohort 4: 1 Dose 30 μg BNT162b2 (B.1.617.2) | Part B - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part C - Cohort 7: 1 Dose of 30 μg BNT162b2 (B.1.1.529) | Part C - Cohort 8: 1 Dose of 30 μg BNT162b2 (Original Vaccine) | Part C - Cohort 9: No Vaccination
Started | 21 | 20 | 20 | 20 | 42 | 17 | 349 | 352 | 361 | 72 | 71 | 35
Completed | 14 | 10 | 15 | 12 | 29 | 13 | 280 | 291 | 299 | 60 | 55 | 30
Not Completed | 7 | 10 | 5 | 8 | 13 | 4 | 69 | 61 | 62 | 12 | 16 | 5
Not completed — Withdrawal of consent | 0 | 0 | 1 | 3 | 3 | 0 | 30 | 9 | 3 | 2 | 5 | 1
Not completed — Lost to Follow-up | 2 | 4 | 2 | 3 | 5 | 2 | 15 | 12 | 38 | 6 | 6 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 7 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 2 | 2 | 4 | 2 | 4 | 22 | 8 | 1 | 3 | 2
Not completed — Protocol Violation | 2 | 3 | 0 | 0 | 1 | 0 | 16 | 18 | 2 | 2 | 2 | 1
Not completed — Not further specified | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Part A and B: Safety Set - All participants who received at least one dose in of IMP. 35 participants were randomized to Part C - Cohort 9. As per protocol, these participants did not receive treatment.
Groups:
- Part A - Cohort 2: 2 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2): Participants received 2 doses of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2) as a single injection one on on Day 1 and on Day 56
- Total: Total of all reporting groups
Arm/Group | Part A - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 2: 2 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 3: 1 Dose of 30 μg BNT162b2 (B.1.1.7) | Part A - Cohort 4: 1 Dose of 30 μg BNT162b2 (B.1.617.2) | Part A - Cohort 5: 1 Dose of 30 μg BNT162b2 (Original Vaccine) | Part A - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part B - Cohort 4: 1 Dose 30 μg BNT162b2 (B.1.617.2) | Part B - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part C - Cohort 7: 1 Dose of 30 μg BNT162b2 (B.1.1.529) | Part C - Cohort 8: 1 Dose of 30 μg BNT162b2 (Original Vaccine) | Part C - Cohort 9: No Vaccination | Total
Number analyzed (Participants) | 21 | 20 | 20 | 20 | 42 | 17 | 349 | 352 | 361 | 72 | 71 | 35 | 1380
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Per the planned analyses, totals were only calculated for participants in Part A , Part B and Part C, respectively.
  years
    Part A: number analyzed (Participants) | 21 | 20 | 20 | 20 | 42 | 17 | 0 | 0 | 0 | 0 | 0 | 0 | 140
    Part A | 35.4 (11.13) | 38.7 (9.79) | 36.0 (11.89) | 39.8 (8.53) | 47.5 (11.10) | 37.1 (11.21) |  |  |  |  |  |  | 40.4 (11.61)
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 349 | 352 | 361 | 0 | 0 | 0 | 1062
    Part B |  |  |  |  |  |  | 48.1 (14.68) | 50.5 (15.27) | 42.1 (15.91) |  |  |  | 46.9 (15.70)
    Part C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 72 | 71 | 35 | 178
    Part C |  |  |  |  |  |  |  |  |  | 41.9 (12.14) | 43.5 (13.57) | 44.5 (11.15) | 43.0 (12.52)
Age, Customized [Count of Participants; unit: Participants]
  18 to 55 years old | 21 | 20 | 20 | 20 | 42 | 17 | 222 | 210 | 242 | 61 | 60 | 31 | 966
  56 to 85 years old | 0 | 0 | 0 | 0 | 0 | 0 | 127 | 142 | 119 | 11 | 11 | 4 | 414
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 10 | 13 | 14 | 11 | 169 | 161 | 204 | 42 | 43 | 25 | 715
  Male | 10 | 8 | 10 | 7 | 28 | 6 | 180 | 191 | 157 | 30 | 28 | 10 | 665
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 4
  Asian | 0 | 1 | 1 | 1 | 4 | 0 | 10 | 6 | 0 | 4 | 4 | 1 | 32
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Black or African American | 0 | 0 | 0 | 0 | 3 | 6 | 50 | 8 | 242 | 4 | 7 | 2 | 322
  White | 20 | 18 | 19 | 19 | 35 | 11 | 258 | 330 | 15 | 62 | 59 | 31 | 877
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 63 | 0 | 0 | 0 | 66
  Multiracial | 0 | 0 | 0 | 0 | 0 | 0 | 30 | 3 | 41 | 0 | 1 | 0 | 75
  Not reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Hispanic or Latino | 7 | 3 | 9 | 1 | 5 | 5 | 30 | 55 | 10 | 12 | 5 | 5 | 147
  Not Hispanic or Latino | 14 | 17 | 11 | 19 | 37 | 12 | 317 | 294 | 348 | 59 | 66 | 30 | 1224
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 3 | 1 | 0 | 0 | 9
Region of Enrollment [Number; unit: participants]
  Turkey | 0 | 0 | 0 | 0 | 0 | 0 | 137 | 0 | 0 | 0 | 0 | 0 | 137
  United States | 21 | 20 | 20 | 20 | 42 | 17 | 134 | 284 | 23 | 62 | 62 | 32 | 737
  South Africa | 0 | 0 | 0 | 0 | 0 | 0 | 78 | 4 | 338 | 0 | 0 | 0 | 420
  Germany | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 64 | 0 | 10 | 9 | 3 | 86
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Per the planned analyses, totals were only calculated for participants in Part A , Part B and Part C, respectively.
  Height was missing for 1 participant in Part A - Cohort 6, 7 participants in Part B - Cohort 1, 13 participants in Part B - Cohort 4 and 3 participants in Part B - Cohort 6. BMI could therefore not be calculated.
  kg/m^2
    Part A: number analyzed (Participants) | 21 | 20 | 20 | 20 | 42 | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 139
    Part A | 27.54 (5.508) | 27.97 (6.840) | 30.09 (6.509) | 29.72 (6.287) | 29.83 (6.722) | 30.82 (8.394) |  |  |  |  |  |  | 29.35 (6.663)
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 342 | 339 | 358 | 0 | 0 | 0 | 1039
    Part B |  |  |  |  |  |  | 28.29 (6.012) | 28.78 (6.202) | 26.30 (8.413) |  |  |  | 27.77 (7.065)
    Part C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 72 | 71 | 35 | 178
    Part C |  |  |  |  |  |  |  |  |  | 29.25 (6.648) | 28.60 (6.581) | 30.23 (5.133) | 29.18 (6.346)

OUTCOME MEASURES:

1. Primary Outcome: All Parts - Percentage of Participants Reporting Local Reactions at the Injection Site (Pain, Tenderness, Erythema/Redness, Induration/Swelling)
Description: Local reactions of any grade are reported. Local reactions were graded using criteria based on the US FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials"; the guidance uses the Grades 1 (mild), 2 (moderate), 3 (severe), and 4 (potentially life-threatening). The reporting of systemic reactions was based on the participant's assessments collected in the electronic diary (e-diary) or mapped from the adverse event case report form from Day 1 to Day 7 after each IMP dose. For Erythema/redness and Induration/swelling, the reported size had to be at least 2.5 cm to be deemed as a local reaction. Local reactions with a size less than 2.5 cm are not included in the analysis. Subjects in Cohort 9 did not receive a vaccination and are not included in this analysis.
Time Frame: from Day 1 to Day 7 after each IMP dose
Population: Reactogenicity set, i.e., all participants included in the Safety Set with any reactogenicity data reported after IMP injection. Per protocol, participants in Part C - Cohort 9 did not receive IMP therefore local reactions were not collected for these participants.
Measure: Count of Participants; unit: Participants
Groups:
- Part A - Cohort 1: 1 Dose of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2); Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2): Participants received 1 dose of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2) as a single injection on Day 1
Arm/Group | Part A - Cohort 1: 1 Dose of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 2: 2 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 3: 1 Dose of 30 μg BNT162b2 (B.1.1.7) | Part A - Cohort 4: 1 Dose of 30 μg BNT162b2 (B.1.617.2) | Part A - Cohort 5: 1 Dose of 30 μg BNT162b2 (Original Vaccine) | Part A - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part B - Cohort 4: 1 Dose 30 μg BNT162b2 (B.1.617.2) | Part B - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part C - Cohort 7: 1 Dose of 30 μg BNT162b2 (B.1.1.529) | Part C - Cohort 8: 1 Dose of 30 μg BNT162b2 (Original Vaccine) | Part C - Cohort 9: No Vaccination
Number analyzed (Participants) | 21 | 20 | 19 | 20 | 40 | 17 | 341 | 348 | 358 | 72 | 70 | 0
Participants
  Any local reaction - Overall | 19 | 20 | 17 | 19 | 37 | 15 | 290 | 310 | 261 | 63 | 61 |
  Pain at the injection site - Overall | 17 | 19 | 14 | 17 | 27 | 13 | 254 | 264 | 247 | 57 | 52 |
  Tenderness - Overall | 18 | 20 | 17 | 18 | 33 | 14 | 220 | 273 | 201 | 55 | 56 |
  Erythema/redness - Overall | 1 | 3 | 1 | 1 | 8 | 1 | 34 | 30 | 47 | 11 | 7 |
  Induration/swelling - Overall | 1 | 3 | 1 | 2 | 10 | 4 | 36 | 30 | 58 | 8 | 5 |
  Any local reaction - After IMP Dose 1: number analyzed (Participants) | 21 | 20 | 19 | 20 | 40 | 16 | 341 | 348 | 347 | 72 | 70 | 0
  Any local reaction - After IMP Dose 1 | 19 | 20 | 17 | 19 | 37 | 12 | 290 | 310 | 213 | 63 | 61 |
  Pain at the injection site - After IMP Dose 1: number analyzed (Participants) | 21 | 20 | 19 | 20 | 40 | 16 | 341 | 348 | 347 | 72 | 70 | 0
  Pain at the injection site - After IMP Dose 1 | 17 | 19 | 14 | 17 | 27 | 10 | 254 | 264 | 194 | 57 | 52 |
  Tenderness - After IMP Dose 1: number analyzed (Participants) | 21 | 20 | 19 | 20 | 40 | 16 | 341 | 348 | 347 | 72 | 70 | 0
  Tenderness - After IMP Dose 1 | 18 | 20 | 17 | 18 | 33 | 12 | 220 | 273 | 133 | 55 | 56 |
  Erythema/redness - After IMP Dose 1: number analyzed (Participants) | 21 | 20 | 19 | 20 | 40 | 16 | 341 | 348 | 347 | 72 | 70 | 0
  Erythema/redness - After IMP Dose 1 | 1 | 3 | 1 | 1 | 8 | 1 | 34 | 30 | 22 | 11 | 7 |
  Induration/swelling - After IMP Dose 1: number analyzed (Participants) | 21 | 20 | 19 | 20 | 40 | 16 | 341 | 348 | 347 | 72 | 70 | 0
  Induration/swelling - After IMP Dose 1 | 1 | 3 | 1 | 2 | 10 | 2 | 36 | 30 | 36 | 8 | 5 |
  Any local reaction - After IMP Dose 2: number analyzed (Participants) | 0 | 14 | 0 | 0 | 0 | 14 | 0 | 0 | 321 | 0 | 0 | 0
  Any local reaction - After IMP Dose 2 |  | 12 |  |  |  | 10 |  |  | 153 |  |  |
  Pain at the injection site - After IMP Dose 2: number analyzed (Participants) | 0 | 14 | 0 | 0 | 0 | 14 | 0 | 0 | 321 | 0 | 0 | 0
  Pain at the injection site - After IMP Dose 2 |  | 11 |  |  |  | 9 |  |  | 142 |  |  |
  Tenderness - After IMP Dose 2: number analyzed (Participants) | 0 | 14 | 0 | 0 | 0 | 14 | 0 | 0 | 321 | 0 | 0 | 0
  Tenderness - After IMP Dose 2 |  | 9 |  |  |  | 10 |  |  | 80 |  |  |
  Erythema/redness - After IMP Dose 2: number analyzed (Participants) | 0 | 14 | 0 | 0 | 0 | 14 | 0 | 0 | 321 | 0 | 0 | 0
  Erythema/redness - After IMP Dose 2 |  | 0 |  |  |  | 0 |  |  | 16 |  |  |
  Induration/swelling - After IMP Dose 2: number analyzed (Participants) | 0 | 14 | 0 | 0 | 0 | 14 | 0 | 0 | 321 | 0 | 0 | 0
  Induration/swelling - After IMP Dose 2 |  | 1 |  |  |  | 0 |  |  | 22 |  |  |
  Any local reaction - After IMP Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 295 | 0 | 0 | 0
  Any local reaction - After IMP Dose 3 |  |  |  |  |  | 8 |  |  | 169 |  |  |
  Pain at the injection site - After IMP Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 295 | 0 | 0 | 0
  Pain at the injection site - After IMP Dose 3 |  |  |  |  |  | 8 |  |  | 153 |  |  |
  Tenderness - After IMP Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 295 | 0 | 0 | 0
  Tenderness - After IMP Dose 3 |  |  |  |  |  | 7 |  |  | 123 |  |  |
  Erythema/redness - After IMP Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 295 | 0 | 0 | 0
  Erythema/redness - After IMP Dose 3 |  |  |  |  |  | 0 |  |  | 19 |  |  |
  Induration/swelling - After IMP Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 295 | 0 | 0 | 0
  Induration/swelling - After IMP Dose 3 |  |  |  |  |  | 3 |  |  | 19 |  |  |

2. Primary Outcome: All Parts - Percentage of Participants Reporting Systemic Events (Fever, Fatigue, Headache, Chills, Vomiting, Nausea, Diarrhea, New or Worsened Muscle Pain, and New or Worsened Joint Pain)
Description: Systemic reactions of any grade are reported. Systemic reactions were graded using criteria based on the guidance given in the US FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials"; the guidance uses the Grades 1 (mild), 2 (moderate), 3 (severe), and 4 (potentially life-threatening). The reporting of systemic reactions was based on the participant's assessments collected in the e-diary or mapped from the adverse event case report form from Day 1 to Day 7 after each IMP dose. For Fever, the reported oral temperature had to be ≥38.0°C to be deemed as a systemic event. Oral temperature less than 38.0°C are not included in the analysis. Subjects in Cohort 9 did not receive a vaccination and are not included in this analysis.
Time Frame: from Day 1 to Day 7 after each IMP dose
Population: Reactogenicity set, i.e., all subjects included in the Safety Set with any reactogenicity data reported after IMP injection. Per protocol, participants in Part C - Cohort 9 did not receive IMP therefore local reactions were not collected for these participants.
Measure: Count of Participants; unit: Participants
Groups:
- Part A - Cohort 2: 2 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2): Participants received 1 dose of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2) as a single injection on Day 1 and one on Day 65
Arm/Group | Part A - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 2: 2 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 3: 1 Dose of 30 μg BNT162b2 (B.1.1.7) | Part A - Cohort 4: 1 Dose of 30 μg BNT162b2 (B.1.617.2) | Part A - Cohort 5: 1 Dose of 30 μg BNT162b2 (Original Vaccine) | Part A - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part B - Cohort 4: 1 Dose 30 μg BNT162b2 (B.1.617.2) | Part B - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part C - Cohort 7: 1 Dose of 30 μg BNT162b2 (B.1.1.529) | Part C - Cohort 8: 1 Dose of 30 μg BNT162b2 (Original Vaccine) | Part C - Cohort 9: No Vaccination
Number analyzed (Participants) | 21 | 20 | 19 | 20 | 40 | 17 | 341 | 347 | 358 | 72 | 70 | 0
Participants
  Any systemic event - Overall | 17 | 20 | 15 | 16 | 33 | 13 | 255 | 267 | 253 | 52 | 55 |
  Fever: Oral temperature of ≥ 38.0℃ - Overall | 4 | 5 | 3 | 2 | 0 | 1 | 32 | 34 | 34 | 1 | 3 |
  Nausea - Overall | 2 | 9 | 4 | 7 | 4 | 4 | 61 | 64 | 93 | 9 | 15 |
  Vomiting - Overall | 0 | 3 | 0 | 1 | 0 | 1 | 8 | 7 | 34 | 1 | 0 |
  Diarrhea - Overall | 2 | 5 | 3 | 2 | 6 | 4 | 19 | 39 | 68 | 8 | 10 |
  Headache - Overall | 15 | 17 | 12 | 8 | 22 | 10 | 160 | 178 | 190 | 32 | 35 |
  Fatigue - Overall | 15 | 19 | 15 | 15 | 30 | 9 | 219 | 220 | 180 | 40 | 44 |
  Chills - Overall | 10 | 13 | 3 | 9 | 13 | 7 | 91 | 115 | 77 | 11 | 14 |
  New or worsened muscle pain - Overall | 10 | 14 | 10 | 8 | 16 | 8 | 123 | 131 | 143 | 20 | 19 |
  New or worsened joint pain - Overall | 6 | 7 | 4 | 4 | 13 | 5 | 87 | 78 | 101 | 9 | 9 |
  Any systemic event - After IMP Dose 1: number analyzed (Participants) | 21 | 20 | 19 | 20 | 40 | 16 | 341 | 347 | 347 | 72 | 70 | 0
  Any systemic event - After IMP Dose 1 | 17 | 18 | 15 | 16 | 33 | 11 | 255 | 267 | 203 | 52 | 55 |
  Fever: Oral temperature of ≥ 38.0℃ - After IMP Dose 1: number analyzed (Participants) | 21 | 20 | 19 | 20 | 40 | 16 | 341 | 347 | 347 | 72 | 70 | 0
  Fever: Oral temperature of ≥ 38.0℃ - After IMP Dose 1 | 4 | 4 | 3 | 2 | 0 | 0 | 32 | 34 | 14 | 1 | 3 |
  Nausea - After IMP Dose 1: number analyzed (Participants) | 21 | 20 | 19 | 20 | 40 | 16 | 341 | 347 | 347 | 72 | 70 | 0
  Nausea - After IMP Dose 1 | 2 | 6 | 4 | 7 | 4 | 3 | 61 | 64 | 58 | 9 | 15 |
  Vomiting - After IMP Dose 1: number analyzed (Participants) | 21 | 20 | 19 | 20 | 40 | 16 | 341 | 347 | 347 | 72 | 70 | 0
  Vomiting - After IMP Dose 1 | 0 | 1 | 0 | 1 | 0 | 1 | 8 | 7 | 22 | 1 | 0 |
  Diarrhea - After IMP Dose 1: number analyzed (Participants) | 21 | 20 | 19 | 20 | 40 | 16 | 341 | 347 | 347 | 72 | 70 | 0
  Diarrhea - After IMP Dose 1 | 2 | 4 | 3 | 2 | 6 | 2 | 19 | 39 | 44 | 8 | 10 |
  Headache - After IMP Dose 1: number analyzed (Participants) | 21 | 20 | 19 | 20 | 40 | 16 | 341 | 347 | 347 | 72 | 70 | 0
  Headache - After IMP Dose 1 | 15 | 16 | 12 | 8 | 22 | 8 | 160 | 178 | 125 | 32 | 35 |
  Fatigue - After IMP Dose 1: number analyzed (Participants) | 21 | 20 | 19 | 20 | 40 | 16 | 341 | 347 | 347 | 72 | 70 | 0
  Fatigue - After IMP Dose 1 | 15 | 17 | 15 | 15 | 30 | 8 | 219 | 220 | 119 | 40 | 44 |
  Chills - After IMP Dose 1: number analyzed (Participants) | 21 | 20 | 19 | 20 | 40 | 16 | 341 | 347 | 347 | 72 | 70 | 0
  Chills - After IMP Dose 1 | 10 | 9 | 3 | 9 | 13 | 3 | 91 | 115 | 43 | 11 | 14 |
  New or worsened muscle pain - After IMP Dose 1: number analyzed (Participants) | 21 | 20 | 19 | 20 | 40 | 16 | 341 | 347 | 347 | 72 | 70 | 0
  New or worsened muscle pain - After IMP Dose 1 | 10 | 12 | 10 | 8 | 16 | 6 | 123 | 131 | 92 | 20 | 19 |
  New or worsened joint pain - After IMP Dose 1: number analyzed (Participants) | 21 | 20 | 19 | 20 | 40 | 16 | 341 | 347 | 347 | 72 | 70 | 0
  New or worsened joint pain - After IMP Dose 1 | 6 | 6 | 4 | 4 | 13 | 3 | 87 | 78 | 68 | 9 | 9 |
  Any systemic event - After IMP Dose 2: number analyzed (Participants) | 0 | 15 | 0 | 0 | 0 | 15 | 0 | 0 | 323 | 0 | 0 | 0
  Any systemic event - After IMP Dose 2 |  | 14 |  |  |  | 9 |  |  | 139 |  |  |
  Fever: Oral temperature of ≥ 38.0℃ - After IMP Dose 2: number analyzed (Participants) | 0 | 15 | 0 | 0 | 0 | 15 | 0 | 0 | 323 | 0 | 0 | 0
  Fever: Oral temperature of ≥ 38.0℃ - After IMP Dose 2 |  | 1 |  |  |  | 1 |  |  | 12 |  |  |
  Nausea - After IMP Dose 2: number analyzed (Participants) | 0 | 15 | 0 | 0 | 0 | 15 | 0 | 0 | 323 | 0 | 0 | 0
  Nausea - After IMP Dose 2 |  | 5 |  |  |  | 2 |  |  | 28 |  |  |
  Vomiting - After IMP Dose 2: number analyzed (Participants) | 0 | 15 | 0 | 0 | 0 | 15 | 0 | 0 | 323 | 0 | 0 | 0
  Vomiting - After IMP Dose 2 |  | 2 |  |  |  | 1 |  |  | 9 |  |  |
  Diarrhea - After IMP Dose 2: number analyzed (Participants) | 0 | 15 | 0 | 0 | 0 | 15 | 0 | 0 | 323 | 0 | 0 | 0
  Diarrhea - After IMP Dose 2 |  | 2 |  |  |  | 2 |  |  | 20 |  |  |
  Headache - After IMP Dose 2: number analyzed (Participants) | 0 | 15 | 0 | 0 | 0 | 15 | 0 | 0 | 323 | 0 | 0 | 0
  Headache - After IMP Dose 2 |  | 11 |  |  |  | 6 |  |  | 88 |  |  |
  Fatigue - After IMP Dose 2: number analyzed (Participants) | 0 | 15 | 0 | 0 | 0 | 15 | 0 | 0 | 323 | 0 | 0 | 0
  Fatigue - After IMP Dose 2 |  | 13 |  |  |  | 6 |  |  | 77 |  |  |
  Chills - After IMP Dose 2: number analyzed (Participants) | 0 | 15 | 0 | 0 | 0 | 15 | 0 | 0 | 323 | 0 | 0 | 0
  Chills - After IMP Dose 2 |  | 6 |  |  |  | 3 |  |  | 29 |  |  |
  New or worsened muscle pain - After IMP Dose 2: number analyzed (Participants) | 0 | 15 | 0 | 0 | 0 | 15 | 0 | 0 | 323 | 0 | 0 | 0
  New or worsened muscle pain - After IMP Dose 2 |  | 9 |  |  |  | 4 |  |  | 61 |  |  |
  New or worsened joint pain - After IMP Dose 2: number analyzed (Participants) | 0 | 15 | 0 | 0 | 0 | 15 | 0 | 0 | 323 | 0 | 0 | 0
  New or worsened joint pain - After IMP Dose 2 |  | 3 |  |  |  | 4 |  |  | 39 |  |  |
  Any systemic event - After IMP Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 295 | 0 | 0 | 0
  Any systemic event - After IMP Dose 3 |  |  |  |  |  | 6 |  |  | 142 |  |  |
  Fever: Oral temperature of ≥ 38.0℃ - After IMP Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 295 | 0 | 0 | 0
  Fever: Oral temperature of ≥ 38.0℃ - After IMP Dose 3 |  |  |  |  |  | 0 |  |  | 13 |  |  |
  Nausea - After IMP Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 295 | 0 | 0 | 0
  Nausea - After IMP Dose 3 |  |  |  |  |  | 1 |  |  | 33 |  |  |
  Vomiting - After IMP Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 295 | 0 | 0 | 0
  Vomiting - After IMP Dose 3 |  |  |  |  |  | 0 |  |  | 12 |  |  |
  Diarrhea - After IMP Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 295 | 0 | 0 | 0
  Diarrhea - After IMP Dose 3 |  |  |  |  |  | 1 |  |  | 22 |  |  |
  Headache - After IMP Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 295 | 0 | 0 | 0
  Headache - After IMP Dose 3 |  |  |  |  |  | 4 |  |  | 104 |  |  |
  Fatigue - After IMP Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 295 | 0 | 0 | 0
  Fatigue - After IMP Dose 3 |  |  |  |  |  | 4 |  |  | 87 |  |  |
  Chills - After IMP Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 295 | 0 | 0 | 0
  Chills - After IMP Dose 3 |  |  |  |  |  | 2 |  |  | 27 |  |  |
  New or worsened muscle pain - After IMP Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 295 | 0 | 0 | 0
  New or worsened muscle pain - After IMP Dose 3 |  |  |  |  |  | 4 |  |  | 54 |  |  |
  New or worsened joint pain - After IMP Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 295 | 0 | 0 | 0
  New or worsened joint pain - After IMP Dose 3 |  |  |  |  |  | 2 |  |  | 28 |  |  |

3. Primary Outcome: All Parts - Percentage of Participants Reporting Adverse Events (AEs)
Description: An AE is defined as TEAE if the event onset date and time is after the first IMP dose (if the event was absent before the first administration of the IMP) or worsened after the first IMP dose (if the event was present before the first administration of the IMP). In the event of an incomplete onset date, the event is considered as treatment-emergent unless the partial onset date information or complete or partial end date confirms the onset date or the event end prior to the first dose of IMP. Percentages for dose 1, dose 2, dose 3 and overall summaries are based upon the number of participants who received the respective IMP dose.
Time Frame: Dose 1 up to 1 month after each dose (all parts)
Population: Safety set, i.e., all participants who received at least one dose of IMP. Per protocol, participants in Part C - Cohort 9 did not receive IMP therefore local reactions were not collected for these participants.
Measure: Number; unit: percentage of participants
Arm/Group | Part A - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 2: 2 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 3: 1 Dose of 30 μg BNT162b2 (B.1.1.7) | Part A - Cohort 4: 1 Dose of 30 μg BNT162b2 (B.1.617.2) | Part A - Cohort 5: 1 Dose of 30 μg BNT162b2 (Original Vaccine) | Part A - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part B - Cohort 4: 1 Dose 30 μg BNT162b2 (B.1.617.2) | Part B - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part C - Cohort 7: 1 Dose of 30 μg BNT162b2 (B.1.1.529) | Part C - Cohort 8: 1 Dose of 30 μg BNT162b2 (Original Vaccine) | Part C - Cohort 9: No Vaccination
Number analyzed (Participants) | 21 | 20 | 20 | 20 | 42 | 17 | 349 | 352 | 361 | 72 | 71 | 0
percentage of participants
  Any AE after IMP Dose 1 | 19.0 | 30.0 | 30.0 | 15.0 | 66.7 | 29.4 | 14.6 | 13.1 | 20.2 | 12.5 | 19.7 |
  Any AE after IMP Dose 2: number analyzed (Participants) | 0 | 20 | 0 | 0 | 0 | 17 | 0 | 0 | 356 | 0 | 0 | 0
  Any AE after IMP Dose 2 |  | 27.8 |  |  |  | 17.6 |  |  | 15.7 |  |  |
  Any AE after IMP Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 315 | 0 | 0 | 0
  Any AE after IMP Dose 3 |  |  |  |  |  | 20.0 |  |  | 15.2 |  |  |

4. Primary Outcome: All Parts - Percentage of Participants Reporting Serious Adverse Events (SAEs)
Description: An SAE was any untoward medical occurrence that, at any dose: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/ incapacity; was a congenital anomaly/birth defect and/or was another important medical event. SAEs from dose 1 up to 6 months post last IMP dose are presented. MedDRA (version 26.1) coding dictionary applied. An SAE is defined as TESAE if the event onset date and time is after the first IMP dose (if the event was absent before the first administration of the IMP) or worsened after the first IMP dose (if the event was present before the first administration of the IMP).
  In the event of an incomplete onset date, the event is considered as treatment-emergent unless the partial onset date information or complete or partial end date confirms the onset date or the event end prior to the first dose of IMP.
Time Frame: Dose 1 up to 6 months after the last dose
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Groups:
- Part A - Cohort 5: 1 Dose of 30 μg BNT162b2 (Orginal Vaccine); Part C - Cohort 8: 1 Dose of 30 μg BNT162b2 (Original Vaccine): Participants received 1 dose of 30 μg BNT162b2 original vaccine on Day 1
Arm/Group | Part A - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 2: 2 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 3: 1 Dose of 30 μg BNT162b2 (B.1.1.7) | Part A - Cohort 4: 1 Dose of 30 μg BNT162b2 (B.1.617.2) | Part A - Cohort 5: 1 Dose of 30 μg BNT162b2 (Orginal Vaccine) | Part A - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part B - Cohort 4: 1 Dose 30 μg BNT162b2 (B.1.617.2) | Part B - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part C - Cohort 7: 1 Dose of 30 μg BNT162b2 (B.1.1.529) | Part C - Cohort 8: 1 Dose of 30 μg BNT162b2 (Original Vaccine) | Part C - Cohort 9: No Vaccination
Number analyzed (Participants) | 21 | 20 | 20 | 20 | 42 | 17 | 349 | 352 | 361 | 72 | 71 | 0
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 1.1 | 1.7 | 3.6 | 0 | 7.0 |

5. Primary Outcome: Part B - GMR of B.1.1.7 NT 1 Month After 1 Dose of BNT162b2 (B.1.1.7 + B.1.617.2) in BNT162b2-experienced Participants to the Reference Strain NT 1 Month After 2 Doses of BNT162b2 in Participants From the Phase III C4591001 (NCT04368728) Trial
Description: GMRs and 2-sided 95% CIs were calculated by exponentiating the difference of least square means and corresponding CIs based on the analysis of logarithmically transformed neutralizing titers using a linear regression model with terms of age, sex, and vaccine group. The overall number of participants analyzed represents the number of participants with valid and determinate assay results for B.1.1.7 and reference strain respectively at the given dose/sampling time point within the specified window. GMR data are presented below as per the primary endpoint defined in the protocol. GMTs for the individual arms (from which GMR was derived) were secondary endpoints and are presented in outcome measure 22.
  GMR = Geometric mean ratio; NT = neutralizing titers
Time Frame: 1 month after booster dose in BNT162-17 participants and 1 month post Dose 2 in participants from the C4591001 (NCT04368728) trial
Population: Immunogenicity Analysis Set, i.e., all eligible randomized/assigned participants who received the trial intervention to which they were randomized or assigned, had a valid and determinate immunogenicity result from the blood sample collected within an appropriate window, and had no other important protocol deviations that could confound immunogenicity data. Includes 332 subjects from C4591001 (NCT04368728).
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratio
Groups:
- BNT162-17 Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) / C4591001 BNT162b2 30 μg: BNT162-17 Part B - Cohort 1 participants received 1 dose of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2) as a single injection on Day 1 and C4591001 (NCT04368728) participants received 2 doses of BNT162b2 30 μg
Arm/Group | BNT162-17 Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) / C4591001 BNT162b2 30 μg
Number analyzed (Participants) | 631
Titer ratio | 8.81 [7.49 to 10.36]

6. Primary Outcome: Part B - GMR of B.1.617.2 NT 1 Month After 1 Dose of BNT162b2 (B.1.1.7 + B.1.617.2) in BNT162b2-experienced Participants to the Reference Strain NT 1 Month After 2 Doses of BNT162b2 in Participants From the Phase III C4591001 (NCT04368728) Trial
Description: GMRs and 2-sided 95% CIs were calculated by exponentiating the difference of least square means and corresponding CIs based on the analysis of logarithmically transformed neutralizing titers using a linear regression model with terms of age, sex, and group. The overall number of participants analyzed represents the number of participants with valid and determinate assay results for B.1.617.2 and reference strain respectively at the given dose/sampling time point within the specified window. GMR data are presented below as per the primary endpoint defined in the protocol. GMTs for the individual arms (from which GMR was derived) were secondary endpoints and are presented in outcome measure 22.
  GMR = Geometric mean ratio; NT = neutralizing titers
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratio
Arm/Group | BNT162-17 Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) / C4591001 BNT162b2 30 μg
Number analyzed (Participants) | 631
Titer ratio | 4.88 [4.19 to 5.68]

7. Primary Outcome: Part B - GMR of B.1.617.2 NT 1 Month After 1 Dose of BNT162b2 (B.1.617.2) in BNT162b2-experienced Participants to the Reference Strain NT 1 Month After 2 Doses of BNT162b2 in Participants From the Phase III C4591001 (NCT04368728) Trial
Description: GMRs and 2-sided 95% CIs were calculated by exponentiating the difference of least square means and corresponding CIs based on the analysis of logarithmically transformed neutralizing titers using a linear regression model with terms of age, sex, and group. The overall number of participants analyzed represents the number of participants with valid and determinate assay results for B.1.617.2 and reference strain respectively at the given dose/sampling time point within the specified window. GMR data are presented below as per the primary endpoint defined in the protocol. GMTs for the individual arms (from which GMR was derived) were secondary endpoints and are presented in outcome measure 24.
Time Frame: as for outcome 5
Population: Immunogenicity Analysis Set, i.e., all eligible randomized/assigned participants who received the trial intervention to which they were randomized or assigned, had a valid and determinate immunogenicity result from the blood sample collected within an appropriate window, and had no other important protocol deviations that could confound immunogenicity data. Includes 320 subjects from C4591001 (NCT04368728).
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratio
Groups:
- BNT162-17 Part B - Cohort 4: 1 Dose 30 μg BNT162b2 (B.1.617.2) / C4591001 BNT162b2 30 μg: BNT162-17 Part B - Cohort 4 participants received 1 dose of 30 μg monovalent vaccine BNT162b2 (B.1.617.2) as a single injection on Day 1 and selected C4591001 (NCT04368728) participants received 2 doses of BNT162b2 30 μg
Arm/Group | BNT162-17 Part B - Cohort 4: 1 Dose 30 μg BNT162b2 (B.1.617.2) / C4591001 BNT162b2 30 μg
Number analyzed (Participants) | 637
Titer ratio | 6.40 [5.47 to 7.48]

8. Primary Outcome: Part B - Difference in Seroresponse (SR) to B.1.1.7 NT 1 Month After 1 Dose of BNT162b2 (B.1.1.7 + B.1.617.2) in BNT162b2-experienced Participants to the Reference Strain NT 1 Month After 2 Doses of BNT162b2 in Participants From C4591001 (NCT04368728)
Description: Seroresponse was defined as a ≥4-fold rise in neutralizing titer from baseline. For subjects with a baseline titer less than the lower limit of quantitation (<LLOQ), seroresponse was defined as a post-vaccination titer of ≥4× LLOQ. Adjusted difference was estimated using minimum risk weights and stratified by sex and age group (18 to 55 years, 56 to 85 years), expressed as a percentage. Associated 2-sided 95% CI based on the Newcombe method with minimum risk weights for the difference in proportions. Difference in seroresponse data are presented below as per the primary endpoint defined in the protocol. Seroresponses for the individual arms (from which the difference was derived) were secondary endpoints and are presented in outcome measure 23.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage difference
Groups:
- BNT162-17 Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) - C4591001 BNT162b2 30 μg: BNT162-17 Part B - Cohort 1 participants received 1 dose of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2) as a single injection on Day 1 and C4591001 (NCT04368728) participants received 2 doses of BNT162b2 30 μg
Arm/Group | BNT162-17 Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) - C4591001 BNT162b2 30 μg
Number analyzed (Participants) | 630
percentage difference | 0.25 [-4.86 to 5.26]

9. Primary Outcome: Part B - Difference in SR to B.1.617.2 NT 1 Month After 1 Dose of BNT162b2 (B.1.1.7 + B.1.617.2) in BNT162b2-experienced Participants to the Reference Strain NT 1 Month After 2 Doses of BNT162b2 in Participants From C4591001 (NCT04368728)
Description: as for outcome 8
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage difference
Arm/Group | BNT162-17 Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) - C4591001 BNT162b2 30 μg
Number analyzed (Participants) | 630
percentage difference | -2.39 [-7.74 to 2.84]

10. Primary Outcome: Part B - Difference in SR to B.1.617.2 NT 1 Month After 1 Dose of BNT162b2 (B.1.617.2) in BNT162b2-experienced Participants to the Reference Strain NT 1 Month After 2 Doses of BNT162b2 in Participants From C4591001 (NCT04368728)
Description: Seroresponse was defined as a ≥4-fold rise in neutralizing titer from baseline. For subjects with a baseline titer less than the lower limit of quantitation (<LLOQ), seroresponse was defined as a post-vaccination titer of ≥4× LLOQ. Adjusted difference was estimated using minimum risk weights and stratified by sex and age group (18 to 55 years, 56 to 85 years), expressed as a percentage. Associated 2-sided 95% CI based on the Newcombe method with minimum risk weights for the difference in proportions. Difference in seroresponse data are presented below as per the primary endpoint defined in the protocol. Seroresponses for the individual arms (from which the difference was derived) were secondary endpoints and are presented in outcome measure 25.
Time Frame: as for outcome 5
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage difference
Groups:
- BNT162-17 Part B - Cohort 4: 1 Dose 30 μg BNT162b2 (B.1.617.2) / C4591001 BNT162b2 30 μg: BNT162-17 Part B - Cohort 4 participants received 1 dose of 30 μg monovalent vaccine BNT162b2 (B.1.617.2) on Day 1 and C4591001 (NCT04368728) participants received 2 doses of BNT162b2 30 μg
Arm/Group | BNT162-17 Part B - Cohort 4: 1 Dose 30 μg BNT162b2 (B.1.617.2) / C4591001 BNT162b2 30 μg
Number analyzed (Participants) | 633
percentage difference | 9.70 [5.68 to 13.97]

11. Primary Outcome: Part B - GMR of B.1.1.7 NT 1 Month After 2 Doses of BNT162b2 (B.1.1.7 + B.1.617.2) in COVID-19 Vaccine-naïve Participants to the Reference Strain NT 1 Month After 2 Doses of BNT162b2 in Participants From the C4591001 (NCT04368728) Trial
Description: Cohort B6 aimed to generate data to support a 2-dose primary regimen of alpha-delta multivalent BNT162b2 vaccine in SARS-CoV-2 naïve, unvaccinated individuals. The population recruited in Cohort B6, while complying with the inclusion criterium of no known history SARS-CoV-2 infection, were retrospectively seropositive for SARS-CoV-2 by planned N-binding antibody assessment of baseline samples. While the cohort was COVID-19 vaccine-naïve, it was not SARS-CoV-2-naïve as needed to match the control group (C4591001/NCT04368728). Procedurally, submission of a protocol amendment was not possible. However, the Statistical Analysis Plan was amended to describe that the non-inferiority analysis could not be performed according to the protocol. Control participants were not selected as planned; therefore, data were not available to calculate the GMR. Available GMT data for the 17 Cohort B6 participants without evidence of infection were analyzed and are presented in Outcome Measure 28.
Time Frame: 1 month
Population: The population recruited in Cohort B6 were retrospectively seropositive for SARS-CoV-2. While the cohort was COVID-19 vaccine-naïve, it was not SARS-CoV-2-naïve as needed to match the control group (C4591001/NCT04368728). Control participants were therefore not selected as planned so data were not available to calculate the GMR. GMT data for the 17 participants without evidence of infection are presented in Outcome Measure 28. Please refer to the outcome measure description for more detail.
Groups:
- BNT162-17 Part B - Cohort 6: 3 Doses 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) / C4591001 BNT162b2 30 μg: BNT162-17 Part B - Cohort 6 participants received 3 doses of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2), as a single injection one on Day 1, one on Day 21 and one approximately 6 months after the second dose. C4591001 (NCT04368728) participants received 1 dose of BNT162b2 30 μg
Arm/Group | BNT162-17 Part B - Cohort 6: 3 Doses 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) / C4591001 BNT162b2 30 μg
Number analyzed (Participants) | 0

12. Primary Outcome: Part B - GMR of B.1.617.2 NT 1 Month After 2 Doses of BNT162b2 (B.1.1.7 + B.1.617.2) in COVID-19 Vaccine-naïve Participants to the Reference Strain NT 1 Month After 2 Doses of BNT162b2 in Participants From the C4591001 (NCT04368728) Trial
Description: Cohort B6 aimed to generate data to support a 2-dose primary regimen of alpha-delta multivalent BNT162b2 vaccine in SARS-CoV-2 naïve, unvaccinated individuals. The population recruited in Cohort B6, while complying with the inclusion criterium of no known history SARS-CoV-2 infection, were retrospectively seropositive for SARS-CoV-2 by planned N-binding antibody assessment of baseline samples. While the cohort was COVID-19 vaccine-naïve, it was not SARS-CoV-2-naïve as needed to match the control group (C4591001/NCT04368728). Procedurally, submission of a protocol amendment was not possible. However, the Statistical Analysis Plan was amended to describe that the non-inferiority analysis could not be performed according to the protocol. Control participants were not selected as planned; therefore, data were not available to calculate the GMR. Available GMT data for the 17 Part B Cohort 6 participants without evidence of infection were analyzed and are presented in Outcome Measure 28.
Time Frame: 1 month
Population: as for outcome 11
Arm/Group | BNT162-17 Part B - Cohort 6: 3 Doses 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) / C4591001 BNT162b2 30 μg
Number analyzed (Participants) | 0

13. Primary Outcome: Part B - The Difference in SR to B.1.1.7 NT 1 Month After 2 Doses of BNT162b2 (B.1.1.7 + B.1.617.2) in COVID-19 Vaccine-naïve Participants to the Reference Strain NT 1 Month After 2 Doses of BNT162b2 in Participants From the C4591001 (NCT04368728) Trial
Description: Cohort B6 aimed to generate data to support a 2-dose primary regimen of alpha-delta multivalent BNT162b2 vaccine in SARS-CoV-2 naïve, unvaccinated individuals. The population recruited in Cohort B6, while complying with the inclusion criterium of no known history SARS-CoV-2 infection, were retrospectively seropositive for SARS-CoV-2 by planned N-binding antibody assessment of baseline samples. While the cohort was COVID-19 vaccine-naïve, it was not SARS-CoV-2-naïve as needed to match the control group (C4591001/NCT04368728). Procedurally, submission of a protocol amendment was not possible. However, the Statistical Analysis Plan was amended to describe that non-inferiority analysis could not be performed according to the protocol. Control participants were not selected as planned; therefore, data were not available to calculate difference in SR. Available SR data for the 17 Part B Cohort 6 participants without evidence of infection were analyzed and presented in Outcome Measure 31.
Time Frame: 1 month
Population: The population recruited in Cohort B6 were retrospectively seropositive for SARS-CoV-2. While the cohort was COVID-19 vaccine-naïve, it was not SARS-CoV-2-naïve as needed to match the control group (C4591001/NCT04368728). Control participants were therefore not selected as planned so data were not available to calculate difference in SR. SR data for 17 participants without evidence of infection are presented in Outcome Measure 31. Please refer to the outcome measure description for more detail.
Arm/Group | BNT162-17 Part B - Cohort 6: 3 Doses 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) / C4591001 BNT162b2 30 μg
Number analyzed (Participants) | 0

14. Primary Outcome: Part B - The Difference in SR to B.1.617.2 NT 1 Month After 2 Doses of BNT162b2 (B.1.1.7 + B.1.617.2) in COVID-19 Vaccine-naïve Participants to the Reference Strain NT 1 Month After 2 Doses of BNT162b2 in Participants From the C4591001 (NCT04368728) Trial
Description: Cohort B6 aimed to generate data to support a 2-dose primary regimen of alpha-delta multivalent BNT162b2 vaccine in SARS-CoV-2 naïve, unvaccinated individuals. The population recruited in Cohort B6, while complying with the inclusion criterium of no known history SARS-CoV-2 infection, were retrospectively seropositive for SARS-CoV-2 by planned N-binding antibody assessment of baseline samples. While the cohort was COVID-19 vaccine-naïve, it was not SARS-CoV-2-naïve as needed to match the control group (C4591001/NCT04368728). Procedurally, submission of a protocol amendment was not possible. However, the Statistical Analysis Plan was amended to describe that the non-inferiority analysis could not be performed according to the protocol. Control participants were not selected as planned; therefore data were not available to calculate difference in SR. Available SR data for the 17 Part B Cohort 6 participants without evidence of infection were analyzed and presented in Outcome Measure 31.
Time Frame: 1 month
Population: as for outcome 13
Arm/Group | BNT162-17 Part B - Cohort 6: 3 Doses 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) / C4591001 BNT162b2 30 μg
Number analyzed (Participants) | 0

15. Primary Outcome: Part B - GMR of Reference Strain NT After One Dose of BNT162b2 (B.1.1.7 + B.1.617.2) in Participants With Evidence of Prior Infection to the Reference Strain NT After 2 Doses of BNT162b2 in Participants Without Evidence of Infection
Description: GMR of reference strain NT 3 weeks (3W) after one dose (PD1) of BNT162b2 (B.1.1.7 + B.1.617.2) in COVID-19 vaccine-naïve participants with evidence of prior infection to the reference strain NT 1 month after two doses of BNT162b2 in participants without evidence of infection (COVID-19 Vaccine-naïve Participants) from the Phase III trial C4591001 (NCT04368728). GMTs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and corresponding CIs (based on the Student t distribution). Assay results below LLOQ were set to 0.5 × LLOQ. GMTs of NTs are presented in the descriptive data section of this outcome measure. GMRs and 2-sided 95% CIs were calculated by exponentiating the difference of LS means and corresponding CIs based on the analysis of logarithmically transformed neutralizing titers using a linear regression model with terms of age, sex, and group. GMR data are presented in the statistical analysis section.
Time Frame: 3 weeks post Dose 1 in BNT162-17 participants and 1 month post Dose 2 in participants from the C4591001 (NCT04368728) trial
Population: Immunogenicity Analysis Set, i.e., all eligible randomized/assigned participants who received the trial intervention to which they were randomized or assigned, had a valid and determinate immunogenicity result from the blood sample collected within an appropriate window, and had no other important protocol deviations that could confound immunogenicity data. Includes 275 participants from C4591001 (NCT04368728).
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- BNT162-17 - C6: 3 Doses 30μg BNT162b2 (B.1.1.7+B.1.617.2) With Evidence of Prior Infection 3W PD1: BNT162-17 Part B - Cohort 6 participants received 3 doses of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2), as a single injection one on Day 1, one on Day 21 and one approximately 6 months after the second dose.
- C4591001 BNT162b2 30 μg Without Evidence of Infection - 1 Month Post-Dose 2: C4591001 (NCT04368728) participants received 2 doses of BNT162b2 30 μg
Arm/Group | BNT162-17 - C6: 3 Doses 30μg BNT162b2 (B.1.1.7+B.1.617.2) With Evidence of Prior Infection 3W PD1 | C4591001 BNT162b2 30 μg Without Evidence of Infection - 1 Month Post-Dose 2
Number analyzed (Participants) | 262 | 275
Titer | 17404.2 [15485.1 to 19561.1] | 1328.1 [1183.1 to 1491.0]
Statistical Analysis 1: Comparison: BNT162-17 - C6: 3 Doses 30μg BNT162b2 (B.1.1.7+B.1.617.2) With Evidence of Prior Infection 3W PD1 vs C4591001 BNT162b2 30 μg Without Evidence of Infection - 1 Month Post-Dose 2; Test type: Non-Inferiority — Noninferiority was declared if the lower bound of the 2-sided 95% CIs for the GMR was greater than 0.67; Geometric mean ratio = 13.12, 95% CI 2-sided [11.14 to 15.45] — GMRs and 2-sided 95% CIs were based on the analysis of logarithmically transformed neutralizing titers using a linear regression model with terms of age, sex, and group

16. Primary Outcome: Part B - The Difference in SRs to the Reference Strain NT in Subjects With Evidence of Prior Infection and to the Reference Strain NT in Participants Without Evidence of Infection (COVID-19 Vaccine-naïve Participants)
Description: The difference in SRs to the reference strain NT 3 weeks after one dose of BNT162b2 (B.1.1.7 + B.1.617.2) in COVID-19 vaccine-naïve participants with evidence of prior infection to the reference strain NT 1 month after two doses of BNT162b2 in participants without evidence of infection from the Phase III trial C4591001 (NCT04368728). SR was defined as achieving a ≥4-fold rise from baseline. If the baseline measurement was below the LLOQ, a post-vaccination assay result ≥4 × LLOQ was considered a SR. SR to the reference strain NTs are presented in the descriptive data section of this outcome measure. Adjusted difference in proportions was estimated using minimum risk weights and stratified by sex and age group (18 to 55 years, 56 to 85 years), expressed as a percentage. 2-Sided CI was based on the Newcombe method with minimum risk weights for the difference in proportions. Difference in SR data are presented in the statistical analysis section.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- BNT162-17 - C6: 3 Doses 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) With Evidence of Prior Infection 3W PD1: BNT162-17 Part B - Cohort 6 participants received 3 doses of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2), as a single injection one on Day 1, one on Day 21 and one approximately 6 months after the second dose.
Arm/Group | BNT162-17 - C6: 3 Doses 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) With Evidence of Prior Infection 3W PD1 | C4591001 BNT162b2 30 μg Without Evidence of Infection - 1 Month Post-Dose 2
Number analyzed (Participants) | 260 | 275
percentage of participants | 85.8 [80.9 to 89.8] | 90.5 [86.5 to 93.7]
Statistical Analysis 1: Comparison: BNT162-17 - C6: 3 Doses 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) With Evidence of Prior Infection 3W PD1 vs C4591001 BNT162b2 30 μg Without Evidence of Infection - 1 Month Post-Dose 2; Test type: Non-Inferiority — Noninferiority was declared if the lower bound of the 2-sided 95% CIs for the difference of percentages was greater than -10%; Difference in Percentages = -4.55, 95% CI 2-sided [-10.04 to 0.83] — Adjusted difference in percentages were estimated using minimum risk weights and stratified by sex and age group

17. Primary Outcome: Part C - GMR of B.1.1.529.1 NT 1 Month After One Dose of BNT162b2 (B.1.1.529.1) in RNA-based COVID-19 Vaccine-experienced Participants With History of SARS-CoV-2 Infection to Those at 1 Month After One Dose of BNT162b2 for Cohorts 7 and 8.
Description: GMRs and 2-sided 95% CIs were calculated by exponentiating the difference of least square means and corresponding CIs based on the analysis of logarithmically transformed neutralizing titers using a linear regression model with terms of age and number of prior doses. The overall number of participants analyzed represents the number of participants with valid and determinate assay results for B.1.1.529.1 at the given dose/sampling time point within the specified window. GMR data are presented below as per the primary endpoint defined in the protocol. GMTs for the individual arms (from which the difference was derived) were secondary endpoints and are presented in outcome measure 32.
Time Frame: 1 month after 1 dose of BNT162b2 or BNT162b2 (B.1.1.529.1)
Population: Immunogenicity Analysis Set, i.e., all eligible randomized/assigned participants who received the trial intervention to which they were randomized or assigned, had a valid and determinate immunogenicity result from the blood sample collected within an appropriate window, and had no other important protocol deviations that could confound immunogenicity data.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratio
Groups:
- Part C - Cohort 7: 1 Dose of 30 μg BNT162b2 / Cohort 8: 1 Dose of 30 μg BNT162b2: Cohort 7 participants received 1 dose of 30 μg monovalent vaccine BNT162b2 (B.1.1.529) on Day 1 and Cohort 8 participants received 1 dose of 30 μg BNT162b2 original vaccine on Day 1
Arm/Group | Part C - Cohort 7: 1 Dose of 30 μg BNT162b2 / Cohort 8: 1 Dose of 30 μg BNT162b2
Number analyzed (Participants) | 121
Titer ratio | 0.94 [0.61 to 1.44]

18. Primary Outcome: Part C - The Difference in SR of B.1.1.529.1 NT 1 Month After One Dose of BNT162b2 (B.1.1.529.1) in RNA-based COVID-19 Vaccine-experienced Participants With History of SARS-CoV-2 Infection to Those at 1 Month After One Dose of BNT162b2 for Cohorts 7 & 8.
Description: SR was defined as a ≥4-fold rise in neutralizing titer from baseline. For participants with a baseline titer less than the lower limit of quantitation (<LLOQ), SR was defined as a post-vaccination titer of ≥4× LLOQ. SR to the reference strain NTs are presented in the descriptive data section of this outcome measure. Adjusted difference was estimated using minimum risk weights and stratified by sex and age group (18 to 55 years, 56 to 85 years), expressed as a percentage. Associated 2-sided 95% CI were based on the Newcombe method with minimum risk weights for the difference in proportions. Difference in SR data are presented in the statistical analysis section.
Time Frame: 1 month after 1 dose of BNT162b2 or BNT162b2 (B.1.1.529.1)
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part C - Cohort 7: 1 Dose of 30 μg BNT162b2 (B.1.1.529): Cohort 7 participants received 1 dose of 30 μg monovalent vaccine BNT162b2 (B.1.1.529) on Day 1
- Part C - Cohort 8: 1 Dose of 30 μg BNT162b2 Original Vaccine: Cohort 8 participants received 1 dose of 30 μg BNT162b2 original vaccine on Day 1
Arm/Group | Part C - Cohort 7: 1 Dose of 30 μg BNT162b2 (B.1.1.529) | Part C - Cohort 8: 1 Dose of 30 μg BNT162b2 Original Vaccine
Number analyzed (Participants) | 64 | 57
percentage of participants | 59.4 [46.4 to 71.5] | 22.8 [12.7 to 35.8]
Statistical Analysis 1: Comparison: Part C - Cohort 7: 1 Dose of 30 μg BNT162b2 (B.1.1.529) vs Part C - Cohort 8: 1 Dose of 30 μg BNT162b2 Original Vaccine; Test type: Other; Difference in Percentages = 36.73, 95% CI 2-sided [19.21 to 51.17] — Adjusted difference was estimated using the minimum risk weights and stratified by sex and age group

19. Secondary Outcome: Part A - Geometric Mean Titer (GMT) at Each Timepoint
Description: For BNT162b2-experienced participants (defined as participants who have previously received two injections of 30 μg BNT162b2). Reference and variant(s) of concern (VOC) specific NT.
  GMTs and 2-sided 95% CIs are calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ are set to 0.5 × LLOQ and above the ULOQ are set to ULOQ.
  Cohorts 1, 3, 4 and 5 received only 1 dose of IMP. Cohort 2 received dose 2 on Day 56 and did not receive dose 3. Cohort 6 received dose 2 on Day 21 and received dose 3 approximately 6 months after dose 2.
Time Frame: Day 1 up to Day 421
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Part A - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 2: 2 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 3: 1 Dose of 30 μg BNT162b2 (B.1.1.7) | Part A - Cohort 4: 1 Dose of 30 μg BNT162b2 (B.1.617.2) | Part A - Cohort 5: 1 Dose of 30 μg BNT162b2 (Orginal Vaccine) | Part A - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2)
Number analyzed (Participants) | 21 | 20 | 20 | 20 | 20 | 17
Titer
  Pre IMP dose 1 - B.1.1.7: number analyzed (Participants) | 19 | 20 | 20 | 20 | 17 | 16
  Pre IMP dose 1 - B.1.1.7 | 18.9 [9.0 to 39.7] | 26.9 [14.5 to 49.9] | 17.4 [9.0 to 33.8] | 48.4 [20.0 to 117.0] | 9.6 [5.2 to 17.8] | 6.9 [4.6 to 10.5]
  1-week post IMP dose 1 - B.1.1.7: number analyzed (Participants) | 15 | 15 | 13 | 15 | 18 | 16
  1-week post IMP dose 1 - B.1.1.7 | 1403.9 [817.9 to 2409.8] | 1340.5 [731.0 to 2458.2] | 1090.8 [701.7 to 1695.5] | 557.2 [365.4 to 849.4] | 307.9 [209.1 to 453.5] | 30.2 [6.8 to 133.1]
  3-weeks post IMP dose 1 - B.1.1.7: number analyzed (Participants) | 18 | 19 | 19 | 20 | 17 | 0
  3-weeks post IMP dose 1 - B.1.1.7 | 1035.7 [659.9 to 1625.5] | 1168.4 [756.8 to 1803.9] | 956.0 [657.3 to 1390.4] | 493.5 [365.0 to 667.3] | 361.6 [223.9 to 584.2] |
  1-month post IMP dose 1 - B.1.1.7: number analyzed (Participants) | 17 | 20 | 19 | 20 | 20 | 0
  1-month post IMP dose 1 - B.1.1.7 | 942.8 [552.6 to 1608.3] | 1004.3 [705.3 to 1430.0] | 1009.8 [697.8 to 1461.3] | 468.5 [308.6 to 711.2] | 314.5 [182.7 to 541.3] |
  6-months post IMP dose 1 - B.1.1.7: number analyzed (Participants) | 16 | 0 | 18 | 19 | 15 | 0
  6-months post IMP dose 1 - B.1.1.7 | 156.6 [62.5 to 392.2] |  | 352.3 [192.4 to 645.3] | 151.5 [68.9 to 333.1] | 85.7 [36.9 to 199.3] |
  12-months post IMP dose 1 - B.1.1.7: number analyzed (Participants) | 12 | 0 | 14 | 11 | 14 | 0
  12-months post IMP dose 1 - B.1.1.7 | 658.8 [385.8 to 1124.7] |  | 463.9 [180.0 to 1195.5] | 241.0 [95.1 to 611.0] | 463.9 [188.0 to 1144.8] |
  Pre IMP dose 2 - B.1.1.7: number analyzed (Participants) | 0 | 18 | 0 | 0 | 0 | 16
  Pre IMP dose 2 - B.1.1.7 |  | 151 [49.1 to 464.5] |  |  |  | 42.7 [12.5 to 145.9]
  1-week post IMP dose 2 - B.1.1.7: number analyzed (Participants) | 0 | 8 | 0 | 0 | 0 | 8
  1-week post IMP dose 2 - B.1.1.7 |  | 987.0 [495.9 to 1964.4] |  |  |  | 207.5 [104.3 to 413.0]
  1-month post IMP dose 2 - B.1.1.7: number analyzed (Participants) | 0 | 18 | 0 | 0 | 0 | 15
  1-month post IMP dose 2 - B.1.1.7 |  | 958.9 [586.3 to 1568.3] |  |  |  | 216.1 [101.7 to 459.0]
  6-months post IMP dose 2 - B.1.1.7: number analyzed (Participants) | 0 | 16 | 0 | 0 | 0 | 0
  6-months post IMP dose 2 - B.1.1.7 |  | 349.0 [166.5 to 731.6] |  |  |  |
  12-months post IMP dose 2 - B.1.1.7: number analyzed (Participants) | 0 | 9 | 0 | 0 | 0 | 0
  12-months post IMP dose 2 - B.1.1.7 |  | 940.6 [480.4 to 1841.7] |  |  |  |
  6-months post IMP dose 2 + pre IMP dose 3 - B.1.1.7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 11
  6-months post IMP dose 2 + pre IMP dose 3 - B.1.1.7 |  |  |  |  |  | 68.3 [21.7 to 215.2]
  1-week post IMP dose 3 - B.1.1.7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7
  1-week post IMP dose 3 - B.1.1.7 |  |  |  |  |  | 640.0 [379.2 to 1080.2]
  1-month post IMP dose 3 - B.1.1.7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8
  1-month post IMP dose 3 - B.1.1.7 |  |  |  |  |  | 562.0 [190.2 to 1660.6]
  12-months post IMP dose 2 + 6-months post IMP dose 3 - B1.1.7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 11
  12-months post IMP dose 2 + 6-months post IMP dose 3 - B1.1.7 |  |  |  |  |  | 351.7 [162.4 to 761.8]
  Pre IMP dose 1 - B.1.617.2: number analyzed (Participants) | 19 | 20 | 20 | 20 | 17 | 16
  Pre IMP dose 1 - B.1.617.2 | 9.0 [4.8 to 16.7] | 8.7 [5.1 to 15.0] | 12.1 [6.4 to 22.8] | 8.7 [6.0 to 12.6] | 9.0 [5.2 to 15.8] | 6.5 [4.7 to 9.0]
  1-week post IMP dose 1 - B.1.617.2: number analyzed (Participants) | 16 | 15 | 13 | 15 | 18 | 16
  1-week post IMP dose 1 - B.1.617.2 | 526.6 [305.8 to 906.9] | 385.0 [255.6 to 579.8] | 517.1 [330.1 to 809.9] | 359.2 [237.3 to 543.7] | 254.0 [162.5 to 396.9] | 27.7 [6.6 to 115.4]
  3-weeks post IMP dose 1 - B.1.617.2: number analyzed (Participants) | 18 | 19 | 19 | 20 | 17 | 0
  3-weeks post IMP dose 1 - B.1.617.2 | 452.5 [283.1 to 723.5] | 384.0 [251.0 to 587.6] | 533.3 [368.0 to 772.7] | 380.5 [265.8 to 544.8] | 221.7 [123.0 to 399.6] |
  1-month post IMP dose 1 - B.1.617.2: number analyzed (Participants) | 17 | 20 | 19 | 20 | 20 | 0
  1-month post IMP dose 1 - B.1.617.2 | 369.1 [209.3 to 650.8] | 303.8 [199.2 to 463.2] | 486.8 [349.2 to 678.6] | 288.4 [199.5 to 417.0] | 207.5 [126.3 to 340.8] |
  6-months post IMP dose 1 - B.1.617.2: number analyzed (Participants) | 16 | 0 | 18 | 19 | 15 | 0
  6-months post IMP dose 1 - B.1.617.2 | 137.5 [51.6 to 366.1] |  | 217.7 [127.9 to 370.5] | 123.9 [55.3 to 277.7] | 35.6 [17.5 to 72.7] |
  12-months post IMP dose 1 - B.1.617.2: number analyzed (Participants) | 12 | 0 | 14 | 11 | 14 | 0
  12-months post IMP dose 1 - B.1.617.2 | 640.0 [293.4 to 1396.1] |  | 199.9 [87.3 to 458.1] | 212.5 [78.3 to 576.2] | 226.3 [92.5 to 553.7] |
  Pre IMP dose 2 - B.1.617.2: number analyzed (Participants) | 0 | 18 | 0 | 0 | 0 | 16
  Pre IMP dose 2 - B.1.617.2 |  | 235.2 [144.0 to 384.1] |  |  |  | 60.4 [18.3 to 199.5]
  1-week post IMP dose 2 - B.1.617.2: number analyzed (Participants) | 0 | 8 | 0 | 0 | 0 | 8
  1-week post IMP dose 2 - B.1.617.2 |  | 515.4 [342.7 to 774.9] |  |  |  | 216.7 [134.6 to 348.7]
  1-month post IMP dose 2 - B.1.617.2: number analyzed (Participants) | 0 | 18 | 0 | 0 | 0 | 15
  1-month post IMP dose 2 - B.1.617.2 |  | 517.8 [366.6 to 731.5] |  |  |  | 320.0 [139.1 to 736.4]
  6-months post IMP dose 2 - B.1.617.2: number analyzed (Participants) | 0 | 16 | 0 | 0 | 0 | 0
  6-months post IMP dose 2 - B.1.617.2 |  | 226.3 [114.9 to 445.6] |  |  |  |
  12-months post IMP dose 2 - B.1.617.2: number analyzed (Participants) | 0 | 9 | 0 | 0 | 0 | 0
  12-months post IMP dose 2 - B.1.617.2 |  | 508.0 [288.7 to 893.9] |  |  |  |
  6-months post IMP dose 2 + pre IMP dose 3 - B.1.617.2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 11
  6-months post IMP dose 2 + pre IMP dose 3 - B.1.617.2 |  |  |  |  |  | 87.9 [26.2 to 294.9]
  1-week post IMP dose 3 - B.1.617.2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7
  1-week post IMP dose 3 - B.1.617.2 |  |  |  |  |  | 819.8 [353.1 to 1903.2]
  1-month post IMP dose 3 - B.1.617.2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8
  1-month post IMP dose 3 - B.1.617.2 |  |  |  |  |  | 640.0 [207.3 to 1976.3]
  12-months post dose 2 + 6-months post dose 3 - B.1.617.2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 11
  12-months post dose 2 + 6-months post dose 3 - B.1.617.2 |  |  |  |  |  | 424.9 [213.3 to 846.5]
  Pre IMP dose 1 - Reference strain: number analyzed (Participants) | 19 | 20 | 20 | 20 | 17 | 16
  Pre IMP dose 1 - Reference strain | 14.9 [8.5 to 26.2] | 18.7 [10.4 to 33.4] | 18.3 [10.1 to 33.3] | 27.8 [16.6 to 46.5] | 14.1 [7.9 to 25.3] | 6.8 [4.6 to 9.9]
  1-week post IMP dose 1 - Reference strain: number analyzed (Participants) | 16 | 15 | 13 | 15 | 18 | 16
  1-week post IMP dose 1 - Reference strain | 812.2 [474.1 to 1391.3] | 519.8 [321.6 to 840.2] | 640.0 [417.4 to 981.4] | 702.0 [432.7 to 1138.7] | 352.3 [238.3 to 521.0] | 25.4 [6.6 to 97.7]
  3-weeks post IMP dose 1 - Reference strain: number analyzed (Participants) | 18 | 19 | 19 | 20 | 17 | 0
  3-weeks post IMP dose 1 - Reference strain | 678.1 [406.0 to 1132.3] | 584.2 [357.5 to 954.8] | 740.6 [495.0 to 1107.8] | 748.0 [500.2 to 1118.6] | 408.7 [262.0 to 637.4] |
  1-month post IMP dose 1 - Reference strain: number analyzed (Participants) | 17 | 20 | 19 | 20 | 20 | 0
  1-month post IMP dose 1 - Reference strain | 589.9 [376.9 to 923.1] | 452.5 [283.5 to 722.4] | 688.4 [467.0 to 1014.9] | 748.0 [469.3 to 1192.3] | 380.5 [232.0 to 624.3] |
  6-months post IMP dose 1 - Reference strain: number analyzed (Participants) | 16 | 0 | 18 | 19 | 15 | 0
  6-months post IMP dose 1 - Reference strain | 163.5 [72.7 to 367.7] |  | 244.4 [143.8 to 415.4] | 101.4 [57.8 to 178.0] | 78.2 [42.2 to 145.0] |
  12-months post IMP dose 1 - Reference strain: number analyzed (Participants) | 12 | 0 | 14 | 11 | 14 | 0
  12-months post IMP dose 1 - Reference strain | 604.1 [311.3 to 1172.1] |  | 380.5 [164.8 to 878.9] | 170.4 [67.6 to 429.5] | 565.5 [244.1 to 1310.2] |
  Pre IMP dose 2 - Reference strain: number analyzed (Participants) | 0 | 18 | 0 | 0 | 0 | 16
  Pre IMP dose 2 - Reference strain |  | 387.9 [227.7 to 660.9] |  |  |  | 37.5 [11.3 to 124.6]
  1-week post IMP dose 2 - Reference strain: number analyzed (Participants) | 0 | 8 | 0 | 0 | 0 | 8
  1-week post IMP dose 2 - Reference strain |  | 697.9 [453.5 to 1074.1] |  |  |  | 95.1 [59.8 to 151.4]
  1-month post IMP dose 2 - Reference strain: number analyzed (Participants) | 0 | 18 | 0 | 0 | 0 | 15
  1-month post IMP dose 2 - Reference strain |  | 665.1 [400.1 to 1105.6] |  |  |  | 136.1 [58.1 to 319.0]
  6-months post IMP dose 2 - Reference strain: number analyzed (Participants) | 0 | 16 | 0 | 0 | 0 | 0
  6-months post IMP dose 2 - Reference strain |  | 334.2 [171.5 to 651.2] |  |  |  |
  12-months post IMP dose 2 - Reference strain: number analyzed (Participants) | 0 | 9 | 0 | 0 | 0 | 0
  12-months post IMP dose 2 - Reference strain |  | 527.9 [263.8 to 1056.2] |  |  |  |
  6-months post IMP dose 2 + pre IMP dose 3 - Reference strain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 11
  6-months post IMP dose 2 + pre IMP dose 3 - Reference strain |  |  |  |  |  | 53.1 [16.4 to 172.4]
  1-week post IMP dose 3 - Reference strain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7
  1-week post IMP dose 3 - Reference strain |  |  |  |  |  | 551.7 [299.8 to 1015.1]
  1-month post IMP dose 3 - Reference strain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8
  1-month post IMP dose 3 - Reference strain |  |  |  |  |  | 493.5 [195.5 to 1245.8]
  12-months post dose 2 + 6-months post dose 3 - Reference strain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 11
  12-months post dose 2 + 6-months post dose 3 - Reference strain |  |  |  |  |  | 205.9 [80.1 to 528.8]

20. Secondary Outcome: Part A - Geometric Mean Fold Rises (GMFR) From Before Vaccination to Each Subsequent Time Point After Vaccination
Description: For BNT162b2-experienced participants (defined as participants who have previously received two injections of 30 μg BNT162b2). Reference and VOC specific NT.
  GMFR is calculated as the mean of the difference of logarithmically transformed neutralization titers or antibody levels (later result minus earlier result) and exponentiating the mean. The associated 2-sided 95% CIs are obtained by constructing CIs using Student's t-distribution for the mean difference on the natural log scale and exponentiating the confidence limits. Assay results below the LLOQ are set to 0.5 × LLOQ and above the ULOQ are set to ULOQ.
  Cohorts 1, 3, 4 and 5 received only 1 dose of IMP. Cohort 2 received dose 2 on Day 56 and did not receive dose 3. Cohort 6 received dose 2 on Day 21 and received dose 3 approximately 6 months after dose 2.
Time Frame: Day 1 to Day 421
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Part A - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 2: 2 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 3: 1 Dose of 30 μg BNT162b2 (B.1.1.7) | Part A - Cohort 4: 1 Dose of 30 μg BNT162b2 (B.1.617.2) | Part A - Cohort 5: 1 Dose of 30 μg BNT162b2 (Orginal Vaccine) | Part A - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2)
Number analyzed (Participants) | 21 | 20 | 20 | 20 | 20 | 17
Fold rise
  1-week post IMP dose 1 - B.1.1.7: number analyzed (Participants) | 15 | 15 | 13 | 15 | 17 | 15
  1-week post IMP dose 1 - B.1.1.7 | 68.6 [30.4 to 155.0] | 78.8 [38.9 to 159.7] | 95.5 [72.0 to 126.5] | 13.0 [5.8 to 28.9] | 31.4 [19.1 to 51.4] | 4.8 [1.2 to 18.9]
  3-weeks post IMP dose 1 - B.1.1.7: number analyzed (Participants) | 18 | 19 | 19 | 20 | 16 | 0
  3-weeks post IMP dose 1 - B.1.1.7 | 52.8 [28.4 to 98.2] | 39.8 [23.3 to 68.0] | 51.4 [30.3 to 87.3] | 10.2 [4.8 to 21.9] | 35.7 [20.6 to 61.6] |
  1-month post IMP dose 1 - B.1.1.7: number analyzed (Participants) | 17 | 20 | 19 | 20 | 17 | 0
  1-month post IMP dose 1 - B.1.1.7 | 48.1 [24.8 to 93.2] | 37.4 [22.8 to 61.4] | 54.3 [31.9 to 92.5] | 9.7 [3.8 to 24.8] | 27.7 [14.0 to 55.2] |
  6-months post IMP dose 1 - B.1.1.7: number analyzed (Participants) | 14 | 0 | 18 | 19 | 12 | 0
  6-months post IMP dose 1 - B.1.1.7 | 7.2 [2.9 to 18.0] |  | 18.7 [8.2 to 42.5] | 2.9 [0.9 to 9.6] | 9.0 [3.7 to 22.0] |
  12-months post IMP dose 1 - B.1.1.7: number analyzed (Participants) | 10 | 0 | 14 | 11 | 11 | 0
  12-months post IMP dose 1 - B.1.1.7 | 21.1 [4.6 to 96.4] |  | 20.5 [6.2 to 68.2] | 4.0 [0.5 to 33.3] | 36.3 [13.8 to 95.5] |
  Pre IMP dose 2 - B.1.1.7: number analyzed (Participants) | 0 | 18 | 0 | 0 | 0 | 16
  Pre IMP dose 2 - B.1.1.7 |  | 6.2 [2.4 to 15.9] |  |  |  | 6.2 [2.2 to 17.4]
  1-week post IMP dose 2 - B.1.1.7: number analyzed (Participants) | 0 | 8 | 0 | 0 | 0 | 8
  1-week post IMP dose 2 - B.1.1.7 |  | 64.0 [37.4 to 109.4] |  |  |  | 41.5 [20.9 to 82.6]
  1-month post IMP dose 2 - B.1.1.7: number analyzed (Participants) | 0 | 18 | 0 | 0 | 0 | 14
  1-month post IMP dose 2 - B.1.1.7 |  | 39.5 [22.2 to 70.6] |  |  |  | 33.6 [17.9 to 63.3]
  6-months post IMP dose 2 - B.1.1.7: number analyzed (Participants) | 0 | 16 | 0 | 0 | 0 | 0
  6-months post IMP dose 2 - B.1.1.7 |  | 15.7 [7.4 to 33.2] |  |  |  |
  12-months post IMP dose 2 - B.1.1.7: number analyzed (Participants) | 0 | 9 | 0 | 0 | 0 | 0
  12-months post IMP dose 2 - B.1.1.7 |  | 22.6 [6.7 to 76.7] |  |  |  |
  6-months post IMP dose 2 + pre IMP dose 3 - B.1.1.7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 11
  6-months post IMP dose 2 + pre IMP dose 3 - B.1.1.7 |  |  |  |  |  | 12.4 [4.3 to 35.8]
  1-week post IMP dose 3 - B.1.1.7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7
  1-week post IMP dose 3 - B.1.1.7 |  |  |  |  |  | 105.0 [76.8 to 143.6]
  1-month post IMP dose 3 - B.1.1.7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7
  1-month post IMP dose 3 - B.1.1.7 |  |  |  |  |  | 82.0 [32.1 to 209.5]
  12-months post dose 2 + 6-months post dose 3 - B.1.1.7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  12-months post dose 2 + 6-months post dose 3 - B.1.1.7 |  |  |  |  |  | 53.8 [25.6 to 113.0]
  1-week post IMP dose 1 - B.1.617.2: number analyzed (Participants) | 16 | 15 | 13 | 15 | 17 | 15
  1-week post IMP dose 1 - B.1.617.2 | 52.7 [28.1 to 98.8] | 64.0 [43.6 to 93.9] | 73.1 [51.1 to 104.6] | 35.9 [21.7 to 59.6] | 27.2 [16.3 to 45.4] | 4.9 [1.2 to 19.5]
  3-weeks post IMP dose 1 - B.1.617.2: number analyzed (Participants) | 18 | 19 | 19 | 20 | 16 | 0
  3-weeks post IMP dose 1 - B.1.617.2 | 48.9 [28.4 to 84.2] | 42.8 [27.6 to 66.5] | 42.1 [26.2 to 67.6] | 43.7 [27.1 to 70.6] | 22.6 [12.3 to 41.7] |
  1-month post IMP dose 1 - B.1.617.2: number analyzed (Participants) | 17 | 20 | 19 | 20 | 17 | 0
  1-month post IMP dose 1 - B.1.617.2 | 40.9 [23.4 to 71.5] | 34.9 [23.5 to 51.7] | 38.4 [22.1 to 66.7] | 33.1 [22.4 to 49.1] | 20.0 [11.7 to 34.2] |
  6-months post IMP dose 1 - B.1.617.2: number analyzed (Participants) | 14 | 0 | 18 | 19 | 12 | 0
  6-months post IMP dose 1 - B.1.617.2 | 13.8 [5.3 to 35.6] |  | 16.3 [8.1 to 32.9] | 14.3 [5.8 to 35.4] | 4.4 [1.9 to 9.9] |
  12-months post IMP dose 1 - B.1.617.2: number analyzed (Participants) | 10 | 0 | 14 | 11 | 11 | 0
  12-months post IMP dose 1 - B.1.617.2 | 42.2 [10.5 to 169.8] |  | 12.8 [4.4 to 37.4] | 21.9 [5.2 to 93.3] | 19.3 [6.9 to 54.0] |
  Pre IMP dose 2 - B.1.617.2: number analyzed (Participants) | 0 | 18 | 0 | 0 | 0 | 16
  Pre IMP dose 2 - B.1.617.2 |  | 27.4 [16.8 to 44.7] |  |  |  | 9.3 [3.2 to 27.5]
  1-week post IMP dose 2 - B.1.617.2: number analyzed (Participants) | 0 | 8 | 0 | 0 | 0 | 8
  1-week post IMP dose 2 - B.1.617.2 |  | 86.7 [53.9 to 139.5] |  |  |  | 43.3 [26.9 to 69.7]
  1-month post IMP dose 2 - B.1.617.2: number analyzed (Participants) | 0 | 18 | 0 | 0 | 0 | 14
  1-month post IMP dose 2 - B.1.617.2 |  | 60.4 [32.9 to 110.8] |  |  |  | 55.2 [24.0 to 126.9]
  6-months post IMP dose 2 - B.1.617.2: number analyzed (Participants) | 0 | 16 | 0 | 0 | 0 | 0
  6-months post IMP dose 2 - B.1.617.2 |  | 26.9 [11.7 to 62.0] |  |  |  |
  12-months post IMP dose 2 - B.1.617.2: number analyzed (Participants) | 0 | 9 | 0 | 0 | 0 | 0
  12-months post IMP dose 2 - B.1.617.2 |  | 34.6 [8.1 to 146.7] |  |  |  |
  6-months post IMP dose 2 + pre IMP dose 3 - B.1.617.2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 11
  6-months post IMP dose 2 + pre IMP dose 3 - B.1.617.2 |  |  |  |  |  | 16.5 [5.0 to 54.5]
  1-week post IMP dose 3 - B.1.617.2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7
  1-week post IMP dose 3 - B.1.617.2 |  |  |  |  |  | 121.8 [63.4 to 233.9]
  1-month post IMP dose 3 - B.1.617.2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7
  1-month post IMP dose 3 - B.1.617.2 |  |  |  |  |  | 86.1 [28.2 to 263.2]
  12-months post dose 2 + 6-months post dose 3 - B.1.617.2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  12-months post dose 2 + 6-months post dose 3 - B.1.617.2 |  |  |  |  |  | 61.8 [30.8 to 124.0]
  1-week post IMP dose 1 - Reference strain: number analyzed (Participants) | 16 | 15 | 13 | 15 | 17 | 15
  1-week post IMP dose 1 - Reference strain | 52.7 [33.3 to 83.2] | 39.4 [21.6 to 71.9] | 50.3 [38.7 to 65.4] | 20.6 [11.0 to 38.7] | 23.1 [15.8 to 33.8] | 4.1 [1.3 to 13.3]
  3-weeks post IMP dose 1 - Reference strain: number analyzed (Participants) | 18 | 19 | 19 | 20 | 16 | 0
  3-weeks post IMP dose 1 - Reference strain | 46.1 [28.1 to 75.8] | 29.2 [18.3 to 46.7] | 37.7 [22.0 to 64.8] | 26.9 [15.6 to 46.3] | 26.3 [16.5 to 42.0] |
  1-month post IMP dose 1 - Reference strain: number analyzed (Participants) | 17 | 20 | 19 | 20 | 17 | 0
  1-month post IMP dose 1 - Reference strain | 40.9 [26.8 to 62.3] | 24.3 [15.0 to 39.1] | 36.4 [20.8 to 63.7] | 26.9 [15.9 to 45.6] | 23.1 [14.7 to 36.3] |
  6-months post IMP dose 1 - Reference strain: number analyzed (Participants) | 14 | 0 | 18 | 19 | 12 | 0
  6-months post IMP dose 1 - Reference strain | 10.5 [5.1 to 21.5] |  | 12.5 [6.1 to 25.4] | 3.7 [1.8 to 7.5] | 5.2 [2.9 to 9.2] |
  12-months post IMP dose 1 - Reference strain: number analyzed (Participants) | 10 | 0 | 14 | 11 | 11 | 0
  12-months post IMP dose 1 - Reference strain | 29.9 [9.2 to 97.1] |  | 17.7 [6.6 to 47.4] | 6.0 [1.4 to 25.1] | 26.5 [11.1 to 63.4] |
  Pre IMP dose 2 - Reference strain: number analyzed (Participants) | 0 | 18 | 0 | 0 | 0 | 16
  Pre IMP dose 2 - Reference strain |  | 21.8 [12.8 to 37.2] |  |  |  | 5.5 [2.0 to 15.1]
  1-week post IMP dose 2 - Reference strain: number analyzed (Participants) | 0 | 8 | 0 | 0 | 0 | 8
  1-week post IMP dose 2 - Reference strain |  | 66.8 [27.7 to 161.5] |  |  |  | 19.0 [12.0 to 30.3]
  1-month post IMP dose 2 - Reference strain: number analyzed (Participants) | 0 | 18 | 0 | 0 | 0 | 14
  1-month post IMP dose 2 - Reference strain |  | 37.3 [21.6 to 64.6] |  |  |  | 21.5 [10.5 to 44.2]
  6-months post IMP dose 2 - Reference strain: number analyzed (Participants) | 0 | 16 | 0 | 0 | 0 | 0
  6-months post IMP dose 2 - Reference strain |  | 18.6 [9.1 to 38.0] |  |  |  |
  12-months post IMP dose 2 - Reference strain: number analyzed (Participants) | 0 | 9 | 0 | 0 | 0 | 0
  12-months post IMP dose 2 - Reference strain |  | 21.0 [5.3 to 83.5] |  |  |  |
  6-months post IMP dose 2 + pre IMP dose 3 - Reference strain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 11
  6-months post IMP dose 2 + pre IMP dose 3 - Reference strain |  |  |  |  |  | 10.0 [3.3 to 30.2]
  1-week post IMP dose 3 - Reference strain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7
  1-week post IMP dose 3 - Reference strain |  |  |  |  |  | 82.0 [52.7 to 127.6]
  1-month post IMP dose 3 - Reference strain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7
  1-month post IMP dose 3 - Reference strain |  |  |  |  |  | 74.2 [34.7 to 158.7]
  12-months post dose 2 + 6-months post dose 3 - Reference strain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  12-months post dose 2 + 6-months post dose 3 - Reference strain |  |  |  |  |  | 32.0 [10.8 to 95.2]

21. Secondary Outcome: Part A - Percentage of Participants Achieving SR in Terms of NT at Each Post Vaccination Time Point
Description: For BNT162b2-experienced participants (defined as participants who have previously received two injections of 30 μg BNT162b2). Reference and VOC specific NT.
  SR is defined as a ≥4-fold rise in neutralizing titer from baseline (pre IMP dose 1). For subjects with a baseline titer less than the LLOQ, SR is defined as a post-vaccination titer of ≥4 × LLOQ. Pre IMP dose 2 is also 2 months post dose 1 for Cohort 2 and 3 weeks post dose 1 for Cohort 6.
  Cohorts 1, 3, 4 and 5 received only 1 dose of IMP. Cohort 2 received dose 2 on Day 56 and did not receive dose 3. Cohort 6 received dose 2 on Day 21 and received dose 3 approximately 6 months after dose 2.
Time Frame: Day 1 to Day 421
Population: as for outcome 17
Measure: Number; unit: Percentage of participants
Arm/Group | Part A - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 2: 2 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 3: 1 Dose of 30 μg BNT162b2 (B.1.1.7) | Part A - Cohort 4: 1 Dose of 30 μg BNT162b2 (B.1.617.2) | Part A - Cohort 5: 1 Dose of 30 μg BNT162b2 (Orginal Vaccine) | Part A - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2)
Number analyzed (Participants) | 21 | 20 | 20 | 20 | 20 | 17
Percentage of participants
  1-week post IMP dose 1 - B.1.1.7: number analyzed (Participants) | 15 | 15 | 13 | 15 | 17 | 15
  1-week post IMP dose 1 - B.1.1.7 | 93.3 | 100 | 100 | 66.7 | 94.1 | 33.3
  3-weeks post IMP dose 1 - B.1.1.7: number analyzed (Participants) | 18 | 19 | 19 | 20 | 16 | 0
  3-weeks post IMP dose 1 - B.1.1.7 | 94.4 | 94.7 | 94.7 | 65.0 | 100.0 |
  1-month post IMP dose 1 - B.1.1.7: number analyzed (Participants) | 17 | 20 | 19 | 20 | 17 | 0
  1-month post IMP dose 1 - B.1.1.7 | 94.1 | 95.0 | 100 | 65.0 | 88.2 |
  6-months post IMP dose 1 - B.1.1.7: number analyzed (Participants) | 14 | 0 | 18 | 19 | 12 | 0
  6-months post IMP dose 1 - B.1.1.7 | 64.3 |  | 83.3 | 47.4 | 75.0 |
  12-months post IMP dose 1 - B.1.1.7: number analyzed (Participants) | 10 | 0 | 14 | 11 | 11 | 0
  12-months post IMP dose 1 - B.1.1.7 | 80.0 |  | 64.3 | 54.5 | 90.9 |
  Pre IMP dose 2 - B.1.1.7: number analyzed (Participants) | 0 | 18 | 0 | 0 | 0 | 16
  Pre IMP dose 2 - B.1.1.7 |  | 61.1 |  |  |  | 43.8
  1-week post IMP dose 2 - B.1.1.7: number analyzed (Participants) | 0 | 8 | 0 | 0 | 0 | 8
  1-week post IMP dose 2 - B.1.1.7 |  | 100 |  |  |  | 100.0
  1-month post IMP dose 2 - B.1.1.7: number analyzed (Participants) | 0 | 18 | 0 | 0 | 0 | 14
  1-month post IMP dose 2 - B.1.1.7 |  | 94.4 |  |  |  | 92.9
  6-months post IMP dose 2 + pre IMP dose 3 - B.1.1.7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 11
  6-months post IMP dose 2 + pre IMP dose 3 - B.1.1.7 |  |  |  |  |  | 63.6
  1-week post IMP dose 3 - B.1.1.7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7
  1-week post IMP dose 3 - B.1.1.7 |  |  |  |  |  | 100.0
  1-month post IMP dose 3 - B.1.1.7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7
  1-month post IMP dose 3 - B.1.1.7 |  |  |  |  |  | 100.0
  6-months post IMP dose 2 - B.1.1.7: number analyzed (Participants) | 0 | 16 | 0 | 0 | 0 | 0
  6-months post IMP dose 2 - B.1.1.7 |  | 87.5 |  |  |  |
  12-months post dose 2 + 6-months post dose 3 - B.1.1.7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  12-months post dose 2 + 6-months post dose 3 - B.1.1.7 |  |  |  |  |  | 100.0
  12-months post IMP dose 2 - B.1.1.7: number analyzed (Participants) | 0 | 9 | 0 | 0 | 0 | 0
  12-months post IMP dose 2 - B.1.1.7 |  | 88.9 |  |  |  |
  1-week post IMP dose 1 - B.1.617.2: number analyzed (Participants) | 16 | 15 | 13 | 15 | 17 | 15
  1-week post IMP dose 1 - B.1.617.2 | 93.8 | 100.0 | 100.0 | 100.0 | 88.2 | 33.3
  3-weeks post IMP dose 1 - B.1.617.2: number analyzed (Participants) | 18 | 19 | 19 | 20 | 16 | 0
  3-weeks post IMP dose 1 - B.1.617.2 | 94.4 | 94.7 | 100.0 | 100.0 | 93.8 |
  1-month post IMP dose 1 - B.1.617.2: number analyzed (Participants) | 17 | 20 | 19 | 20 | 17 | 0
  1-month post IMP dose 1 - B.1.617.2 | 100.0 | 95.0 | 94.7 | 100.0 | 88.2 |
  6-months post IMP dose 1 - B.1.617.2: number analyzed (Participants) | 14 | 0 | 18 | 19 | 12 | 0
  6-months post IMP dose 1 - B.1.617.2 | 78.6 |  | 88.9 | 73.7 | 58.3 |
  12-months post IMP dose 1 - B.1.617.2: number analyzed (Participants) | 10 | 0 | 14 | 11 | 11 | 0
  12-months post IMP dose 1 - B.1.617.2 | 90.0 |  | 57.1 | 81.8 | 81.8 |
  Pre IMP dose 2 - B.1.617.2: number analyzed (Participants) | 0 | 18 | 0 | 0 | 0 | 16
  Pre IMP dose 2 - B.1.617.2 |  | 94.4 |  |  |  | 56.3
  1-week post IMP dose 2 - B.1.617.2: number analyzed (Participants) | 0 | 8 | 0 | 0 | 0 | 8
  1-week post IMP dose 2 - B.1.617.2 |  | 100 |  |  |  | 100
  1-month post IMP dose 2 - B.1.617.2: number analyzed (Participants) | 0 | 18 | 0 | 0 | 0 | 14
  1-month post IMP dose 2 - B.1.617.2 |  | 94.4 |  |  |  | 92.9
  6-months post IMP dose 2 + pre IMP dose 3 - B.1.617.2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 11
  6-months post IMP dose 2 + pre IMP dose 3 - B.1.617.2 |  |  |  |  |  | 72.7
  1-week post IMP dose 3 - B.1.617.2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7
  1-week post IMP dose 3 - B.1.617.2 |  |  |  |  |  | 100.0
  1-month post IMP dose 3 - B.1.617.2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7
  1-month post IMP dose 3 - B.1.617.2 |  |  |  |  |  | 100.0
  6-months post IMP dose 2 - B.1.617.2: number analyzed (Participants) | 0 | 16 | 0 | 0 | 0 | 0
  6-months post IMP dose 2 - B.1.617.2 |  | 81.3 |  |  |  |
  12-months post dose 2 + 6-months post dose 3 - B.1.617.2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  12-months post dose 2 + 6-months post dose 3 - B.1.617.2 |  |  |  |  |  | 100
  12-months post IMP dose 2 - B.1.617.2: number analyzed (Participants) | 0 | 9 | 0 | 0 | 0 | 0
  12-months post IMP dose 2 - B.1.617.2 |  | 88.9 |  |  |  |
  1-week post IMP dose 1 - Reference strain: number analyzed (Participants) | 16 | 15 | 13 | 15 | 17 | 15
  1-week post IMP dose 1 - Reference strain | 100 | 100.0 | 100.0 | 86.7 | 94.1 | 33.3
  3-weeks post IMP dose 1 - Reference strain: number analyzed (Participants) | 18 | 19 | 19 | 20 | 16 | 0
  3-weeks post IMP dose 1 - Reference strain | 100 | 100.0 | 94.7 | 95.0 | 100.0 |
  1-month post IMP dose 1 - Reference strain: number analyzed (Participants) | 17 | 20 | 19 | 20 | 17 | 0
  1-month post IMP dose 1 - Reference strain | 100 | 95.0 | 94.7 | 95.0 | 100.0 |
  6-months post IMP dose 1 - Reference strain: number analyzed (Participants) | 14 | 0 | 18 | 19 | 12 | 0
  6-months post IMP dose 1 - Reference strain | 64.3 |  | 83.3 | 36.8 | 58.3 |
  12-months post IMP dose 1 - Reference strain: number analyzed (Participants) | 10 | 0 | 14 | 11 | 11 | 0
  12-months post IMP dose 1 - Reference strain | 90.0 |  | 85.7 | 54.5 | 90.9 |
  Pre IMP dose 2 - Reference strain: number analyzed (Participants) | 0 | 18 | 0 | 0 | 0 | 16
  Pre IMP dose 2 - Reference strain |  | 94.4 |  |  |  | 43.8
  1-week post IMP dose 2 - Reference strain: number analyzed (Participants) | 0 | 8 | 0 | 0 | 0 | 8
  1-week post IMP dose 2 - Reference strain |  | 100.0 |  |  |  | 100.0
  1-month post IMP dose 2 - Reference strain: number analyzed (Participants) | 0 | 18 | 0 | 0 | 0 | 14
  1-month post IMP dose 2 - Reference strain |  | 100.0 |  |  |  | 85.7
  6-months post IMP dose 2 + pre IMP dose 3 - Reference strain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 11
  6-months post IMP dose 2 + pre IMP dose 3 - Reference strain |  |  |  |  |  | 54.5
  1-week post IMP dose 3 - Reference strain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7
  1-week post IMP dose 3 - Reference strain |  |  |  |  |  | 100.0
  1-month post IMP dose 3 - Reference strain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7
  1-month post IMP dose 3 - Reference strain |  |  |  |  |  | 100.0
  6-months post IMP dose 2 - Reference strain: number analyzed (Participants) | 0 | 16 | 0 | 0 | 0 | 0
  6-months post IMP dose 2 - Reference strain |  | 93.8 |  |  |  |
  12-months post dose 2 + 6-months post dose 3 - Reference strain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10
  12-months post dose 2 + 6-months post dose 3 - Reference strain |  |  |  |  |  | 100.0
  12-months post IMP dose 2 - Reference strain: number analyzed (Participants) | 0 | 9 | 0 | 0 | 0 | 0
  12-months post IMP dose 2 - Reference strain |  | 88.9 |  |  |  |

22. Secondary Outcome: Part B - GMT of VOCs and Reference Strains in Part B Cohort 1 and Control
Description: GMTs of VOCs (B.1.1.7 and B.1.617.2) and reference strain 1 month after 1 dose of BNT162 (B.1.1.7+B.1.167.2) in participants from Part B Cohort 1 of the BNT162-17 trial (BNT162b2-experienced participants), and reference strain 1 month after 2 doses of BNT162b2 in selected participants from the Phase III C4591001 (NCT04368728) trial.
  GMTs and 2-sided 95% CIs are calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ are set to 0.5 × LLOQ and above the ULOQ are set to ULOQ.
Time Frame: as for outcome 5
Population: Immunogenicity Analysis Set Immunogenicity Analysis Set, i.e., all eligible randomized/assigned participants who received the trial intervention to which they were randomized or assigned, had a valid and determinate immunogenicity result from the blood sample collected within an appropriate window, and had no other important protocol deviations that could confound immunogenicity data. Includes 332 subjects from C4591001 (NCT04368728).
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- BNT162-17 Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2): Participants received 1 dose of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2) as a single injection on Day 1
- C4591001 BNT162b2 30 μg: Participants had previously received two injections of 30 μg BNT162b2 at least 6 months after the second BNT162b2 dose
Arm/Group | BNT162-17 Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | C4591001 BNT162b2 30 μg
Number analyzed (Participants) | 299 | 332
Titer
  B.1.1.7 | 996.5 [880.3 to 1128.0] | 74.7 [66.1 to 84.3]
  B.1.617.2 | 552.4 [495.2 to 616.2] | 65.2 [57.5 to 74.0]
  Reference strain | 947.0 [846.4 to 1059.5] | 113.3 [101.4 to 126.5]

23. Secondary Outcome: Part B - SR of of VOCs and Reference Strains in Part B Cohort 1 and Control
Description: Percentage of participants achieving SR at 1 month after 1 dose of BNT162b2 (B.1.1.7 + B.1.617.2) in BNT162b2-experienced participants (Cohort 1) and 1 month after 2 doses of BNT162b2 primary series (participants from C4591001 [NCT04368728]). SR is defined as a ≥4-fold rise in neutralizing titer from baseline (pre IMP dose 1). For participants with a baseline titer less than the LLOQ, SR is defined as a post-vaccination titer of ≥4 × LLOQ.
Time Frame: 1 month after Dose 1 in BNT162-17 participants and 1 month post Dose 2 in participants from the C4591001 (NCT04368728) trial
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2): Participants in Part B - Cohort 1 received 1 dose of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2) as a single injection on Day 1
Arm/Group | Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | C4591001 BNT162b2 30 μg
Number analyzed (Participants) | 298 | 332
Percentage of participants
  B.1.1.7 | 88.6 [84.4 to 92.0] | 76.2 [71.3 to 80.7]
  B.1.617.2 | 85.9 [81.4 to 89.6] | 74.4 [69.3 to 79.0]
  Reference strain | 89.6 [85.6 to 92.8] | 88.3 [84.3 to 91.5]

24. Secondary Outcome: Part B - GMT of VOCs and Reference Strains in Part B Cohort 4 and Control
Description: GMTs of VOCs (B.1.617.2) and reference strain 1 month after 1 dose of BNT162 (B.1.167.2) in participants from Part B Cohort 4 of the BNT162-17 trial (BNT162b2-experienced participants), and 1 month after 2 doses of BNT162b2 in selected participants from the Phase III C4591001 (NCT04368728) trial.
  GMTs and 2-sided 95% CIs are calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ are set to 0.5 × LLOQ and above the ULOQ are set to ULOQ.
Time Frame: as for outcome 5
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- Part B - Cohort 4 - 1 Dose 30 μg BNT162b2 (B.1.617.2): Participants in Part B - Cohort 4 received 1 dose of 30 μg monovalent vaccine BNT162b2 (B.1.617.2) on Day 1
Arm/Group | Part B - Cohort 4 - 1 Dose 30 μg BNT162b2 (B.1.617.2) | C4591001 BNT162b2 30 μg
Number analyzed (Participants) | 317 | 320
Titer
  B.1.1.7 | 972.8 [875.3 to 1081.1] | 78.6 [69.6 to 88.8]
  B.1.617.2 | 730.5 [654.5 to 815.3] | 71.2 [62.7 to 80.8]
  Reference strain | 1005.3 [900.3 to 1122.5] | 113.0 [100.5 to 127.1]

25. Secondary Outcome: Part B - SR of of VOCs and Reference Strains in Part B Cohort 4 and Control
Description: Percentage of participants achieving SR at 1 month after 1 dose of BNT162b2 (B.1.617.2) in BNT162b2-experienced subjects (Part B - Cohort 4) and 1 month after 2 doses of BNT162b2 primary series (participants from C4591001 [NCT04368728]). SR is defined as a ≥4-fold rise in neutralizing titer from baseline (pre IMP dose 1). For participants with a baseline titer less than the LLOQ, SR is defined as a post-vaccination titer of ≥4 × LLOQ.
Time Frame: as for outcome 23
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B - Cohort 4 - 1 Dose 30 μg BNT162b2 (B.1.617.2) | C4591001 BNT162b2 30 μg
Number analyzed (Participants) | 313 | 320
Percentage of participants
  B.1.1.7 | 96.5 [93.8 to 98.2] | 78.4 [73.5 to 82.8]
  B.1.617.2 | 97.4 [95.0 to 98.9] | 77.5 [72.5 to 82.0]
  Reference strain | 98.1 [95.9 to 99.3] | 87.5 [83.4 to 90.9]

26. Secondary Outcome: Part B - GMT of VOCs and Reference Strain in Part B Cohort 6 1 Month After Dose 2 and 1 Month After Dose 3
Description: GMTs of VOCs and reference strain NT 1 month after dose 2 and dose 3 of BNT162b2 (B.1.1.7 + B.1.617.2) (Part B - Cohort 6). GMTs and 2-sided 95% CIs are calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ are set to 0.5 × LLOQ and above the ULOQ are set to ULOQ.
Time Frame: 1 month after Dose 2 and 1 month after Dose 3
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- Part B - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.6172): Participants in Part B - Cohort 6 received 3 doses of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2), as a single injection one on Day 1, one on Day 21 and one approximately 6 months after the second dose.
Arm/Group | Part B - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.6172)
Number analyzed (Participants) | 359
Titer
  1 month post IMP dose 2 - B.1.1.7: number analyzed (Participants) | 282
  1 month post IMP dose 2 - B.1.1.7 | 832.5 [718.2 to 965.0]
  1 month post IMP dose 3 - B.1.1.7: number analyzed (Participants) | 290
  1 month post IMP dose 3 - B.1.1.7 | 942.6 [836.4 to 1062.4]
  1 month post IMP dose 2 - B.1.617.2: number analyzed (Participants) | 282
  1 month post IMP dose 2 - B.1.617.2 | 1184.6 [1015.5 to 1381.9]
  1 month post IMP dose 3 - B.1.617.2: number analyzed (Participants) | 290
  1 month post IMP dose 3 - B.1.617.2 | 1270.9 [1130.2 to 1429.0]
  1 month post IMP dose 2 - Reference strain: number analyzed (Participants) | 282
  1 month post IMP dose 2 - Reference strain | 697.5 [594.0 to 819.1]
  1 month post IMP dose 3 - Reference strain: number analyzed (Participants) | 290
  1 month post IMP dose 3 - Reference strain | 830.5 [736.3 to 936.8]

27. Secondary Outcome: Part B - Cohort 6 - Percentages With SRs to VOCs (B.1.1.7, B.1.617.2) and Reference Strain
Description: Percentage of participants achieving SR to VOCs (B.1.1.7, B.1.617.2) and reference strain at 1 month after dose 2 and dose 3 of BNT162b2 (B.1.1.7 + B.1.617.2) (Part B - Cohort 6).
  SR is defined as a ≥4-fold rise in neutralizing titer from baseline (pre IMP dose 1). For participants with a baseline titer less than the LLOQ, SR is defined as a post vaccination titer of ≥4 × LLOQ. Pre IMP dose 2 is also 3 weeks post dose 1 for Cohort 6.
Time Frame: 1 month after Dose 2 and 1 month after Dose 3
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.6172)
Number analyzed (Participants) | 359
Percentage of participants
  1 month post IMP dose 2 - B.1.1.7: number analyzed (Participants) | 280
  1 month post IMP dose 2 - B.1.1.7 | 86.8 [82.2 to 90.5]
  1 month post IMP dose 3 - B.1.1.7: number analyzed (Participants) | 287
  1 month post IMP dose 3 - B.1.1.7 | 83.6 [78.8 to 87.7]
  1 month post IMP dose 2 - B.1.617.2: number analyzed (Participants) | 280
  1 month post IMP dose 2 - B.1.617.2 | 88.9 [84.7 to 92.4]
  1 month post IMP dose 3 - B.1.617.2: number analyzed (Participants) | 287
  1 month post IMP dose 3 - B.1.617.2 | 87.1 [82.7 to 90.8]
  1 month post IMP dose 2 - Reference strain: number analyzed (Participants) | 280
  1 month post IMP dose 2 - Reference strain | 87.5 [83.0 to 91.1]
  1 month post IMP dose 3 - Reference strain: number analyzed (Participants) | 287
  1 month post IMP dose 3 - Reference strain | 89.5 [85.4 to 92.8]

28. Secondary Outcome: Part B - GMTs of VOC in COVID-19 Vaccine-naïve Participants With and Without Evidence of Prior Infection in Part B C6 (1 and 2 Primary Doses Respectively) and in BNT162b2-Experienced Participants Without Evidence of Infection in Part B C1 (1 Booster Dose)
Description: GMTs of VOC specific NTs (B.1.1.7, B.1.617.2, B.1.1.529.5 [Omicron BA.5]) 3 weeks after one dose of BNT162b2 (B.1.1.7 + B.1.617.2) in COVID-19 vaccine-naïve participants with evidence of prior infection (Cohort 6), 1 month after two doses of BNT162b2 (B.1.1.7 + B.1.617.2) in COVID-19 vaccine-naïve participants without evidence of infection (Cohort 6), and 1 month after one booster dose of BNT162b2 (B.1.1.7 + B.1.617.2) in BNT162b2-experienced participants without evidence of infection (Cohort 1). GMTs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5 × LLOQ; assay results above the ULOQ were set to ULOQ.
Time Frame: Day 1 up to 1 month after 1 booster dose in Part B Cohort 1 without evidence of infection, up to 1 month after 2 doses in Part B Cohort 6 without evidence of infection and up to 3 weeks after 1 dose in Part B Cohort 6 with evidence of prior infection
Population: Immunogenicity Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- Part B - Cohort 6: BNT162b2 With Evidence of Prior Infection; Part B - Cohort 6: BNT162b2 Without Evidence of Infection: Participants received 3 doses of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2), as a single injection one on Day 1, one on Day 21 and one approximately 6 months after the second dose
- Part B - Cohort 1: BNT162b2 Without Evidence of Infection: Participants received 1 dose of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2) as a single injection on Day 1
Arm/Group | Part B - Cohort 6: BNT162b2 With Evidence of Prior Infection | Part B - Cohort 6: BNT162b2 Without Evidence of Infection | Part B - Cohort 1: BNT162b2 Without Evidence of Infection
Number analyzed (Participants) | 142 | 17 | 136
Titer
  SARS-CoV-2 neutralization assay - B.1.1.7 | 1045.3 [853.1 to 1280.8] | 180.8 [91.8 to 356.3] | 749.5 [621.1 to 904.6]
  SARS-CoV-2 neutralization assay - B.1.617.2 | 859.9 [693.4 to 1066.4] | 62.6 [30.9 to 127.0] | 466.6 [401.8 to 541.9]
  SARS-CoV-2 neutralization assay - B.1.1.529.5 | 229.3 [191.7 to 274.4] | 10.2 [5.7 to 18.3] | 80.8 [66.9 to 97.6]

29. Secondary Outcome: Part B - GMRs of VOC in COVID-19 Vaccine-naïve Participants With and Without Evidence of Prior Infection (1 and 2 Primary Doses Respectively) and in BNT162b2-Experienced Participants Without Evidence of Infection (1 Booster Dose)
Description: GMR of VOC specific NTs (B.1.1.7, B.1.617.2, B.1.1.529.5 [Omicron BA.5]) 3 weeks after one dose of BNT162b2 (B.1.1.7 + B.1.617.2) in COVID-19 vaccine-naïve participants with evidence of prior infection (Cohort 6) to the VOCs NTs 1 month after two doses of BNT162b2 (B.1.1.7 + B.1.617.2) in participants without evidence of infection (Cohort 6), and to the VOCs NTs 1 month after one booster dose of BNT162b2 (B.1.1.7 + B.1.617.2) in BNT162b2-experienced participants without evidence of infection (Cohort 1). GMRs and 2-sided 95% CIs were calculated by exponentiating the difference of the LS means and corresponding CIs based on the analysis of logarithmically transformed neutralizing titers using a linear regression model with terms of age, sex, and group. A separate model was fit for each comparison. Assay results below the LLOQ were set to 0.5 × LLOQ; assay results above the ULOQ were set to ULOQ.
Time Frame: Day 1 to Day 29
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratio
Groups:
- Part B - Cohort 6 With Prior Infection / Cohort 6 Without Prior Infection: Participants in Cohort 6 with or without evidence of prior infection received 3 doses of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2), as a single injection one on Day 1, one on Day 21 and one approximately 6 months after the second dose
- Part B - Cohort 6 With Prior Infection / Cohort 1 Without Prior Infection: Participants in Cohort 6 with evidence of infection received 3 doses of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2), as a single injection one on Day 1, one on Day 21 and one approximately 6 months after the second dose. Participants in Cohort 1 without prior evidence of infection received 1 dose of 30 μg multivalent vaccine BNT162b2 (B.1.1.7 + B.1.617.2) as a single injection on Day 1
Arm/Group | Part B - Cohort 6 With Prior Infection / Cohort 6 Without Prior Infection | Part B - Cohort 6 With Prior Infection / Cohort 1 Without Prior Infection
Number analyzed (Participants) | 159 | 278
Titer ratio
  SARS-CoV-2 neutralization assay - B.1.1.7 | 7.66 [4.09 to 14.33] | 1.46 [1.10 to 1.93]
  SARS-CoV-2 neutralization assay - B.1.617.2 | 15.43 [7.87 to 30.28] | 1.88 [1.44 to 2.45]
  SARS-CoV-2 neutralization assay - B.1.1.529.5 | 29.86 [17.31 to 51.49] | 2.94 [2.26 to 3.82]

30. Secondary Outcome: Part B - Difference in SRs to VOCs in COVID-19 Vaccine-naïve Participants With and Without Evidence of Prior Infection (1 and 2 Primary Doses Respectively) and in BNT162b2-Experienced Participants Without Evidence of Infection (1 Booster Dose)
Description: The difference in SRs to VOC specific NTs (B.1.1.7, B.1.617.2, B.1.1.529.5 [Omicron BA.5]) 3 weeks after one dose of BNT162b2 (B.1.1.7 + B.1.617.2) in COVID-19 vaccine-naïve participants with evidence of prior infection (Cohort 6) to those 1 month after two doses of BNT162b2 (B.1.1.7 + B.1.617.2) in participants without evidence of infection (Cohort 6), and to those 1 month after one booster dose of BNT162b2 (B.1.1.7 + B.1.617.2) in BNT162b2-experienced participants without evidence of infection (Cohort 1). Adjusted difference in proportions estimated using minimum risk weights and stratified by sex and age group (18 to 55 years, 56 to 85 years), expressed as a percentage. 2-Sided CI based on the Newcombe method stratified by sex and age group (18 to 55 years, 56 to 85 years) with minimum risk weights for the difference in proportions.
Time Frame: Day 1 to Day 29
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage difference
Arm/Group | Part B - Cohort 6 With Prior Infection / Cohort 6 Without Prior Infection | Part B - Cohort 6 With Prior Infection / Cohort 1 Without Prior Infection
Number analyzed (Participants) | 159 | 278
Percentage difference
  SARS-CoV-2 neutralization assay - B.1.1.7 | 6.95 [-9.69 to 32.17] | -9.75 [-16.43 to -3.24]
  SARS-CoV-2 neutralization assay - B.1.617.2 | 20.90 [-0.62 to 46.52] | -6.56 [-13.03 to -0.37]
  SARS-CoV-2 neutralization assay - B.1.1.529.5 | 81.47 [54.28 to 90.07] | 6.67 [-2.06 to 15.42]

31. Secondary Outcome: Part B - SR of VOC in COVID-19 Vaccine-naïve Participants With and Without Evidence of Prior Infection (1 and 2 Primary Doses Respectively) and in BNT162b2-Experienced Participants Without Evidence of Infection (1 Booster Dose)
Description: SRs of VOC specific NTs (B.1.1.7, B.1.617.2, B.1.1.529.5 [Omicron BA.5]) 3 weeks after one dose of BNT162b2 (B.1.1.7 + B.1.617.2) in COVID-19 vaccine-naïve participants with evidence of prior infection (Cohort 6) 1 month after two doses of BNT162b2 (B.1.1.7 + B.1.617.2) in participants without evidence of infection (Cohort 6), and 1 month after one booster dose of BNT162b2 (B.1.1.7 + B.1.617.2) in BNT162b2-experienced participants without evidence of infection (Cohort 1). Seroresponse was defined as achieving a ≥4-fold rise from baseline. If the baseline measurement was below the LLOQ, a postvaccination assay result ≥4 × LLOQ was considered a seroresponse.
Time Frame: 3 weeks after one dose in participants with evidence of prior infection (Cohort 6), 1 month after two doses in participants without evidence of infection (Cohort 6), and 1 month after one booster dose (Cohort 1)
Population: as for outcome 17
Measure: Number (97.5% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B - Cohort 6: BNT162b2 With Evidence of Prior Infection | Part B - Cohort 6: BNT162b2 Without Evidence of Infection | Part B - Cohort 1: BNT162b2 Without Evidence of Infection
Number analyzed (Participants) | 142 | 17 | 136
Percentage of participants
  SARS-CoV-2 neutralization assay - B.1.1.7 | 87.3 [80.7 to 92.3] | 76.5 [50.1 to 93.2] | 97.1 [92.6 to 99.2]
  SARS-CoV-2 neutralization assay - B.1.617.2 | 89.4 [83.2 to 94.0] | 58.8 [32.9 to 81.6] | 96.3 [91.6 to 98.8]
  SARS-CoV-2 neutralization assay - B.1.1.529.5 | 87.3 [80.7 to 92.3] | 11.8 [1.5 to 36.4] | 80.1 [72.4 to 86.5]

32. Secondary Outcome: Part C - GMT - B.1.1.529.1 in RNA Based COVID-19 Vaccine-experienced Participants With History of SARS-CoV-2 Infection
Description: VOC NT in RNA-based COVID-19 vaccine-experienced participants with history of SARS-CoV-2 infection at baseline and 7 days, 1 month, and 3 months after the trial start for Cohorts 7, 8, and 9, and 6 and 12 months after the trial start for Cohorts 7 and 8.
  GMTs and 2-sided 95% CIs are calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ are set to 0.5 × LLOQ and above the ULOQ are set to ULOQ. Number of subjects with valid and determinate assay results for the specified variant at the given dose/sampling time point. No vaccination was given to Cohort 9 participants within 3 months after Visit 1. The term "post IMP" does not apply for Cohort 9 since no IMP was given, but blood was collected at the same timepoints post randomization.
Time Frame: Day 1 to Day 360
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- Part C - Cohort 7: 1 Dose of 30 μg BNT162b2 (B.1.1.529.1): Participants in Part C - Cohort 7 received 1 dose of 30 μg monovalent vaccine BNT162b2 (B.1.1.529.1) on Day 1
- Part C - Cohort 8: 1 Dose of 30 μg BNT162b2 (Original Vaccine): Participants in Part C - Cohort 8 received 1 dose of 30 μg BNT162b2 original vaccine on Day 1
- Part C - Cohort 9: No Vaccination: No vaccination was given to Part C - Cohort 9 participants within 3 months after Visit 1. After the 3-month follow-up period, participants in Cohort 9 were to be offered a BNT162b2 vaccination, depending on the epidemiological situation, local regulatory authority recommendations, and/or variant vaccine authorization status.
  35 participants were randomized to Part C - Cohort 9. As per protocol, these participants did not receive treatment.
Arm/Group | Part C - Cohort 7: 1 Dose of 30 μg BNT162b2 (B.1.1.529.1) | Part C - Cohort 8: 1 Dose of 30 μg BNT162b2 (Original Vaccine) | Part C - Cohort 9: No Vaccination
Number analyzed (Participants) | 68 | 59 | 28
Titer
  Baseline | 169.2 [124.4 to 230.2] | 388.5 [262.0 to 575.9] | 164.0 [96.1 to 280.0]
  1-week post IMP Dose 1: number analyzed (Participants) | 56 | 51 | 26
  1-week post IMP Dose 1 | 751.7 [571.5 to 988.9] | 768.9 [550.0 to 1074.9] | 211.7 [122.5 to 365.9]
  1-month post IMP Dose 1: number analyzed (Participants) | 64 | 57 | 26
  1-month post IMP Dose 1 | 748.8 [572.0 to 980.3] | 801.5 [569.8 to 1127.4] | 180.4 [106.7 to 305.0]
  3-months post IMP Dose 1: number analyzed (Participants) | 60 | 49 | 22
  3-months post IMP Dose 1 | 590.3 [433.6 to 803.6] | 571.5 [411.5 to 793.8] | 143.3 [86.7 to 236.9]
  6-months post IMP Dose 1: number analyzed (Participants) | 59 | 51 | 0
  6-months post IMP Dose 1 | 289.6 [210.7 to 397.9] | 356.8 [266.9 to 476.8] |
  12-months post IMP Dose 1: number analyzed (Participants) | 55 | 46 | 0
  12-months post IMP Dose 1 | 197.0 [142.5 to 272.3] | 180.5 [135.9 to 239.8] |

ADVERSE EVENTS:
Time Frame: AEs: From Dose 1 to 1 Month after each dose; SAEs: From Dose 1 up to end of study, i.e., up to 18 months.
Description: 35 participants were randomized to Part C - Cohort 9. As per protocol, these participants did not receive treatment and therefore adverse event data were not collected for these participants
Arm/Group | Part A - Cohort 1: 1 Dose of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 2: 2 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part A - Cohort 3: 1 Dose of 30 μg BNT162b2 (B.1.1.7) | Part A - Cohort 4: 1 Dose of 30 μg BNT162b2 (B.1.617.2) | Part A - Cohort 5: 1 Dose of 30 μg BNT162b2 (Original Vaccine) | Part A - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part B - Cohort 4: 1 Dose 30 μg BNT162b2 (B.1.617.2) | Part B - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) | Part C - Cohort 7: 1 Dose of 30 μg BNT162b2 (B.1.1.529) | Part C - Cohort 8: 1 Dose of 30 μg BNT162b2 (Original Vaccine)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 0/20 | 0/20 | 0/42 | 0/17 | 1/349 | 0/352 | 2/361 | 0/72 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/20 | 1/20 | 0/20 | 0/42 | 0/17 | 6/349 | 9/352 | 13/361 | 0/72 | 5/71
Other Adverse Events (participants affected / at risk) | 2/21 | 7/20 | 4/20 | 0/20 | 27/42 | 6/17 | 26/349 | 0/352 | 39/361 | 4/72 | 5/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - Cohort 1: 1 Dose of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) (N=21) | Part A - Cohort 2: 2 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) (N=20) | Part A - Cohort 3: 1 Dose of 30 μg BNT162b2 (B.1.1.7) (N=20) | Part A - Cohort 4: 1 Dose of 30 μg BNT162b2 (B.1.617.2) (N=20) | Part A - Cohort 5: 1 Dose of 30 μg BNT162b2 (Original Vaccine) (N=42) | Part A - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) (N=17) | Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) (N=349) | Part B - Cohort 4: 1 Dose 30 μg BNT162b2 (B.1.617.2) (N=352) | Part B - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) (N=361) | Part C - Cohort 7: 1 Dose of 30 μg BNT162b2 (B.1.1.529) (N=72) | Part C - Cohort 8: 1 Dose of 30 μg BNT162b2 (Original Vaccine) (N=71)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cor pulmonale (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localized infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Physical assault (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - Cohort 1: 1 Dose of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) (N=21) | Part A - Cohort 2: 2 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) (N=20) | Part A - Cohort 3: 1 Dose of 30 μg BNT162b2 (B.1.1.7) (N=20) | Part A - Cohort 4: 1 Dose of 30 μg BNT162b2 (B.1.617.2) (N=20) | Part A - Cohort 5: 1 Dose of 30 μg BNT162b2 (Original Vaccine) (N=42) | Part A - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) (N=17) | Part B - Cohort 1: 1 Dose 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) (N=349) | Part B - Cohort 4: 1 Dose 30 μg BNT162b2 (B.1.617.2) (N=352) | Part B - Cohort 6: 3 Doses of 30 μg BNT162b2 (B.1.1.7 + B.1.617.2) (N=361) | Part C - Cohort 7: 1 Dose of 30 μg BNT162b2 (B.1.1.529) (N=72) | Part C - Cohort 8: 1 Dose of 30 μg BNT162b2 (Original Vaccine) (N=71)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 4 (7) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 26 (26) | 0 (0) | 39 (42) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Product administration error (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 22 (22) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators respectively trial sites shall not publish or refer to in writing or orally, in whole or in part, any data, information or materials generated from the study and the services, without the prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/81/NCT05004181/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT05004181/SAP_001.pdf